CLINICAL TRIAL: NCT00999518
Title: A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE RANGING STUDY EVALUATING THE EFFICACY AND SAFETY OF TANEZUMAB FOR THE TREATMENT OF MODERATE TO SEVERE PAIN ASSOCIATED WITH INTERSTITIAL CYSTITIS/ PAINFUL BLADDER SYNDROME (IC/PBS).
Brief Title: A Study To Investigate Tanezumab In Patients With Interstitial Cystitis/ Painful Bladder Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091035; 2009-014597-17 (EudraCT Number)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Cystitis, Interstitial
Keywords: Randomized double blind placebo-controlled parallel-group dose-range finding interstitial cystitis efficacy pain urinary symptoms safety
MeSH Terms: conditions — Cystitis, Interstitial | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental)
  Interventions: Biological: Tanezumab
- Group 2 (Experimental)
  Interventions: Biological: Tanezumab
- Group 3 (Experimental)
  Interventions: Biological: Tanezumab
- Group 4 (Experimental)
  Interventions: Biological: Tanezumab
- Group 5 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tanezumab — 1 mg dose given subcutaneously twice at an 8-week interval.
  Arms: Group 1
Biological: Tanezumab — 2.5 mg dose given subcutaneously twice at an 8-week interval.
  Arms: Group 2
Biological: Tanezumab — 10 mg dose given subcutaneously twice at an 8-week interval.
  Arms: Group 3
Biological: Tanezumab — 20 mg dose given subcutaneously twice at an 8-week interval.
  Arms: Group 4
Other: Placebo — Placebo dose given subcutaneously twice at an 8-week interval.
  Arms: Group 5

SUMMARY:
In a previous study in patients with interstitial cystitis/ painful bladder syndrome (IC/PBS), tanezumab has shown to be efficacious in relieving the pain associated with IC/PBS, as well as some effect on reducing urinary urgency. Only one dose was studied, and tanezumab was well tolerated. In this study, the hypothesis being tested is that tanezumab will show efficacy at several doses on reducing pain with sufficient tolerability. Tanezumab's safety will also be assessed at different dose levels

DETAILED DESCRIPTION:
This study was terminated on 16 November 2010 following a US FDA partial clinical hold for the tanezumab interstitial cystitis clinical study announced on 19 July 2010 for potential safety issues, and following a pre-planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with interstitial cystitis/ painful bladder syndrome for more than 6 months with moderate to severe pain and a micturition frequency greater than 7 per day.
* Patients who have been on stable oral medicines for interstitial cystitis/ painful bladder syndrome for at least 3 months. Other therapies might need to be stopped.

Exclusion Criteria:

* Patients on certain recent treatments for interstitial cystitis/ painful bladder syndrome.
* Body mass index (BMI) of >39 kg/m2.
* History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG-fusion protein.
* Patients with peripheral neuropathy.
* Patients with Type I or type II diabetes mellitus who have an HbA1c > 8.0%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2010-01-22 (Actual); Primary Completion 2010-11-17 (Actual); Study Completion 2011-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (171):
- United States (122):
  - Alabama Orthopaedic Clinic, Mobile, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Canyon State Urology, Glendale, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Urology Specialists, Ltd., Phoenix, Arizona
  - Central Arizona Urologists, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Precision Trials, LLC, Phoenix, Arizona
  - Valley Radiologists (x-ray only), Phoenix, Arizona
  - Valley Urologic Associates, Phoenix, Arizona
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - Radiology Limited (x-ray only), Tucson, Arizona
  - Arizona Urologic Specialists, Tucson, Arizona
  - Access Medical Imaging, Beverly Hills, California
  - Urology Associates of Central California, Fresno, California
  - Citrus Valley Medical Research Inc., Glendora, California
  - Atlantic Urology Medical Group, Long Beach, California
  - Institute for Advanced Urology, Los Angeles, California
  - Tri Valley Urology Group, Murrieta, California
  - Valley Neurology, Murrieta, California
  - Liberty Pacific Medical Imaging, Signal Hill, California
  - Boulder Medical Center, PC, Boulder, Colorado
  - Longmont Clinic, PC, Longmont, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Grove Hill Clinical Research, New Britain, Connecticut
  - Urology Center of Grove Hill, New Britain, Connecticut
  - Brian J. Hines, MD, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Diagnostic Imaging (radiology only), Dover, Delaware
  - Urology Associates of Dover, Dover, Delaware
  - Visions Clinical Research, Boynton Beach, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University Urologists, Lake Worth, Florida
  - Specialists in Urology, Naples, Florida
  - Advanced Urology Associates, New Port Richey, Florida
  - Excel Medical Imaging, New Port Richey, Florida
  - Urology Specialists of West Florida, New Port Richey, Florida
  - Advanced Imaging Center Incorporated, Ocala, Florida
  - Ocala Urology Specialists, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Gateway Radiology (x-rays only), Pinellas Park, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Advanced Research Institute Incorporated, Trinity, Florida
  - Midtown Imaging, West Palm Beach, Florida
  - Atlanta Medical Research Institute, LLC, Alpharetta, Georgia
  - Northside Hospital Radiology Services (x-ray only), Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - MRI Imaging of Georgia, Atlanta, Georgia
  - MRI Imaging Of Georgia, Atlanta, Georgia
  - Georgia Urology, Decatur, Georgia
  - Deaconess Clinic Downtown Research Institute, Evansville, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Deaconess Clinic Gateway Health Center Research Institute, Newburgh, Indiana
  - American Health Network (X-Ray only), Noblesville, Indiana
  - Urology of Indiana, LLC, Noblesville, Indiana
  - The Iowa Clinic, Medical Imaging, West Des Moines, Iowa
  - The Iowa Clinic, Urology, West Des Moines, Iowa
  - Regional Urology, LLC, Shreveport, Louisiana
  - Anne Arundel Diagnostics Imaging, Annapolis, Maryland
  - Anne Arundel Urology, PA, Annapolis, Maryland
  - Alpha Clinical Research, Brighton, Massachusetts
  - Genesis Clinical Research and Consulting, Fall River, Massachusetts
  - Grand Rapids Women's Health dba Female Pelvic Medicine and Urogynecology Institute of Michigan, Grand Rapids, Michigan
  - HealthCare Midwest, Kalamazoo, Michigan
  - Rheumatology PC, Kalamazoo, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Beaumont Hospitals - Royal Oak, Royal Oak, Michigan
  - Michigan Institute of Urology, P.C., Troy, Michigan
  - CRL Imaging Southdale (x-rays only), Edina, Minnesota
  - Medical Advanced Pain Specialists Applied Research Center Incorporated, Edina, Minnesota
  - Southeast Urology Network, Southaven, Mississippi
  - Family Health Care Center (X-Ray), Lincoln, Nebraska
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Capital Region Urological Surgeons, Albany, New York
  - Benedictine Hospital, Kingston, New York
  - Hudson Valley Urology, PC, Kingston, New York
  - University Urology Associates, New York, New York
  - DRA Imaging, PC (X-Rays Only), Poughkeepsie, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Rochester, Department of Urology, Rochester, New York
  - Crescent Medical Research, Salisbury, North Carolina
  - Salisbury Urological Clinic, Salisbury, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Tri-State Urologic Services PSC, Inc. dba The Urology Group, Cincinnati, Ohio
  - Central Ohio Urology Group, Cofumbus, Ohio
  - Columbus Urology Research, LLC, Columbus, Ohio
  - Premier Urology, Westerville, Ohio
  - Legacy Clinical Research, LLC, Oklahoma City, Oklahoma
  - Planned Parenthood of Arkansas and Eastern Oklahoma, Tulsa, Oklahoma
  - Oklahoma State University, Tulsa, Oklahoma
  - Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Jeanes Hospital, Philadelphia, Pennsylvania
  - Matrix Research, LLC, Greer, South Carolina
  - The Urology Group, Greer, South Carolina
  - Bristol Urological Associates, PC, Bristol, Tennessee
  - TriCities Medical Research, Bristol, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - University Urology, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - The Neurology Clinic, Memphis, Tennessee
  - Southeast Urology Network, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Access Clinical Trials, Inc (ACT), Nashville, Tennessee
  - Center for Urological Treatment, Nashville, Tennessee
  - Diagnostic Health, Nashville, Tennessee
  - Swan and Brennan, Incorporated, Nashville, Tennessee
  - The Center for Reproductive Health, Nashville, Tennessee
  - Mobley Research Center, Houston, Texas
  - Advances In Health, Inc., Houston, Texas
  - St. Luke's Diagnostic and Treatment Center Kirby Glen, Houston, Texas
  - Centex Research, Inc., Houston, Texas
  - Rocky Mountain Neurological Associates, Murray, Utah
  - Salt Lake Surgical Center, Murray, Utah
  - Salt Lake Regional Medical Center (X-rays only), Salt Lake City, Utah
  - Salt Lake Research, PLLC, Salt Lake City, Utah
  - Western Urological Clinic, PC, Salt Lake City, Utah
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - Urology Northwest, Mountlake Terrace, Washington
  - Marc Kirschner, MD, Seattle, Washington
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Gasthuisberg, Leuven
- Canada (8):
  - The Gateway 2, Abbotsford, British Columbia
  - The Male/Female Health and Research Centre, Royal Court Medical Centre, Barrie, Ontario
  - Centre for Applied Urological Research, Kingston, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Urology Associates / Urologic Medical Research, Kitchener, Ontario
  - Anthony Skehan Medicine Professional Corporation, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Kouvolan Laakariasema, Kouvola, Finland
- Hong Kong (2):
  - Department of Obstetrics & Gynaecology, Prince of Wales Hospital The Chinese University of Hong Kong, Shatin, NEW Territories
  - Department of Surgery, The Chinese University of Hong Kong, Shatin
- Japan (4):
  - Harasanshin Hospital, Urology, Fukuoka, Fukuoka
  - Kyoto City Hospital, Urology, Nakagyo-ku, Kyoto-shi, Kyoto
  - Tokyo Women's Medical University Medical Center East, Arakawa-ku, Tokyo
  - Tokyo University Hospital, Bunkyo-ku, Tokyo
- Poland (5):
  - SPZOZ Wojewodzki Szpital Zespolony im. Jedrzeja Sniadeckiego, Oddzial Urologii, Bialystok
  - Conti Medica Sp. z o.o., Warsaw
  - Spoldzielnia Pracy Specjalistow Radiologow, Warsaw
  - NZOZ Centrum Medyczne Wola, Warsaw
  - Szpital Kliniczny Dzieciatka Jezus, Centrum Leczenia Obrazen, Warsaw
- Romania (3):
  - Dinu Uromedica SCM, Bucharest, Sector 4
  - Spitalul Clinic Prof. Dr. Th. Burghele, Bucharest
  - Centrul Medical Sf. Pantelimon, Pantelimon
- Russia (5):
  - Federal State Institution Scientific Research Institute of Urology of Rosmedtechnology, Moscow
  - Urology of Rosmedtechnology, Moscow
  - Saint-Petersburg State Healthcare Institution City Hospital # 15/Department of Urology, Saint Petersburg
  - SEIHPE St. Petersburg State Medical University n.a.I.P. Pavlov Roszdrava, Saint Petersburg
  - SEIHPE St. Petersburg State Medical University n.a.I.P. Pavlov Roszdrava/Chair of Urology, Saint Petersburg
- Slovakia (3):
  - Martinska fakultna nemocnica, Martin
  - Univerzitna nemocnica Martin, Martin
  - MILAB s.r.o., Prešov
- South Korea (4):
  - Department of Urology, Asan Medical Center, University of Ulsan, Songpa-gu, Seoul
  - Department of Urology, Seoul National University Hospital, Seoul
  - Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Department of Urology, Korea University Anam Hospital, Seoul
- Spain (3):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Clinica Del Remei - Instituto Medico Tecnologico, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
- Sweden (3):
  - Kliniska provningsenheten, Gothenburg
  - Medicinsk Rontgen (x-ray only), Malmo
  - Center for Lakemedelsprovning Malmo, Malmo
- Taiwan (4):
  - Chang Gung Medical Foundation - Kaohsiung/Department of Surgery, Koahsiung Hsien
  - Taichung Hospital, Department of Health, Executive Yuan, Taichung
  - Taipei Veterans General Hospital (X-Ray Only), Taipei
  - Taipei Veterans General Hospital/Department of Surgery, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091035&StudyName=A%20Study%20To%20Investigate%20Tanezumab%20In%20Patients%20With%20Interstitial%20Cystitis/%20Painful%20Bladder%20Syndrome

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) subcutaneous injection at Day 1 and Week 8. Participants were followed up to Week 24.
- Tanezumab 1 mg: Tanezumab (RN624 or PF-04383119) 1 milligram (mg) subcutaneous injection at Day 1 and Week 8. Participants were followed up to Week 24.
- Tanezumab 2.5 mg: Tanezumab (RN624 or PF-04383119) 2.5 mg subcutaneous injection at Day 1 and Week 8. Participants were followed up to Week 24.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg subcutaneous injection at Day 1 and Week 8. Participants were followed up to Week 24.
- Tanezumab 20 mg: Tanezumab (RN624 or PF-04383119) 20 mg subcutaneous injection at Day 1 and Week 8. Participants were followed up to Week 24.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Started | 43 | 42 | 39 | 40 | 41
Treated | 42 | 41 | 37 | 40 | 40
Completed | 19 | 17 | 17 | 18 | 17
Not Completed | 24 | 25 | 22 | 22 | 24
Not completed — Adverse Event | 1 | 6 | 3 | 1 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 1
Not completed — Did not meet entrance criteria | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 10 | 6 | 5 | 5 | 9
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 5 | 4 | 10 | 6 | 1
Not completed — Other | 5 | 7 | 1 | 4 | 5
Not completed — Randomized but not Treated | 1 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who had received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg | Total
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (13.5) | 45.2 (14.9) | 47.2 (13.1) | 51.3 (14.5) | 45.3 (14.2) | 48.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 31 | 36 | 32 | 170
  Male | 4 | 8 | 6 | 4 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Average Daily Pain Score at Week 8
Description: Average daily pain score was defined as the mean of the last 7 daily diary pain ratings prior to each assessment time point. Participants rated their average bladder pain due to interstitial cystitis/painful bladder syndrome (IC/PBS) over the past 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 = no bladder pain to 10 = worst possible bladder pain.
Time Frame: Baseline, Week 8
Population: ITT analysis set included all randomized participants who had received at least 1 dose of study medication. Here 'number analyzed' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
units on a scale
  Baseline | 5.38 (1.259) | 5.72 (1.337) | 6.01 (1.381) | 5.76 (1.669) | 6.08 (1.288)
  Change at Week 8: number analyzed (Participants) | 38 | 32 | 31 | 34 | 34
  Change at Week 8 | -1.21 (1.682) | -1.16 (1.760) | -1.49 (2.502) | -1.60 (2.175) | -1.57 (1.610)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 1 mg; The 3 parameter E max dose-response model, including baseline as a covariate, was fitted to estimate mean difference (tanezumab minus placebo) and associated 95% confidence interval (CI); Test type: Superiority or Other; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.40 to 0.35]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5 mg; The 3 parameter E max dose-response model, including baseline as a covariate, was fitted to estimate mean difference (tanezumab minus placebo) and associated 95% CI; Test type: Superiority or Other; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.80 to 0.68]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-1.15 to 0.83]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.93 to 0.47]

2. Secondary Outcome: Change From Baseline in Mean Average Daily Pain Score at Week 1, 2, 3, 4, 5, 6, 7, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: ITT analysis set included all randomized participants who had received at least 1 dose of study medication. Here 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'Number analyzed' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 36 | 39 | 40
units on a scale
  Change at Week 1 | -0.45 (1.100) | -0.45 (0.997) | -0.83 (1.715) | -0.39 (0.821) | -0.43 (1.055)
  Change at Week 2: number analyzed (Participants) | 41 | 41 | 36 | 39 | 40
  Change at Week 2 | -0.91 (1.296) | -0.55 (1.151) | -1.07 (2.039) | -0.73 (1.450) | -0.99 (1.273)
  Change at Week 3: number analyzed (Participants) | 41 | 39 | 35 | 39 | 39
  Change at Week 3 | -1.14 (1.521) | -0.90 (1.642) | -1.09 (2.135) | -1.10 (1.590) | -1.17 (1.283)
  Change at Week 4: number analyzed (Participants) | 40 | 36 | 34 | 37 | 39
  Change at Week 4 | -1.06 (1.559) | -1.14 (1.797) | -1.50 (2.153) | -1.41 (1.789) | -1.41 (1.640)
  Change at Week 5: number analyzed (Participants) | 39 | 36 | 31 | 36 | 37
  Change at Week 5 | -1.18 (1.576) | -1.09 (1.686) | -1.51 (2.121) | -1.52 (2.063) | -1.56 (1.456)
  Change at Week 6: number analyzed (Participants) | 38 | 35 | 30 | 35 | 36
  Change at Week 6 | -0.97 (1.650) | -1.43 (1.815) | -1.69 (2.084) | -1.42 (2.074) | -1.47 (1.537)
  Change at Week 7: number analyzed (Participants) | 40 | 31 | 30 | 34 | 36
  Change at Week 7 | -1.18 (1.814) | -1.53 (1.894) | -1.67 (2.308) | -1.61 (2.131) | -1.66 (1.770)
  Change at Week 9: number analyzed (Participants) | 37 | 29 | 28 | 31 | 31
  Change at Week 9 | -1.31 (1.774) | -1.62 (1.844) | -1.68 (2.439) | -1.74 (2.219) | -1.74 (1.485)
  Change at Week 10: number analyzed (Participants) | 33 | 26 | 25 | 28 | 30
  Change at Week 10 | -1.42 (1.881) | -1.37 (1.930) | -1.95 (2.628) | -1.61 (1.822) | -1.98 (1.779)
  Change at Week 11: number analyzed (Participants) | 32 | 28 | 23 | 29 | 29
  Change at Week 11 | -1.53 (1.770) | -1.41 (1.961) | -2.10 (2.504) | -1.85 (2.502) | -1.95 (1.884)
  Change at Week 12: number analyzed (Participants) | 31 | 27 | 24 | 28 | 29
  Change at Week 12 | -1.62 (1.598) | -1.28 (1.768) | -1.93 (2.177) | -1.84 (2.517) | -1.94 (1.630)
  Change at Week 13: number analyzed (Participants) | 33 | 26 | 23 | 25 | 29
  Change at Week 13 | -1.58 (1.751) | -1.47 (1.944) | -2.05 (2.129) | -1.83 (2.374) | -2.16 (1.678)
  Change at Week 14: number analyzed (Participants) | 32 | 24 | 23 | 24 | 27
  Change at Week 14 | -1.56 (1.882) | -1.41 (2.195) | -1.86 (1.988) | -1.68 (2.355) | -1.85 (1.760)
  Change at Week 15: number analyzed (Participants) | 28 | 24 | 22 | 25 | 23
  Change at Week 15 | -1.50 (1.785) | -1.81 (1.710) | -2.00 (1.959) | -1.68 (2.399) | -2.03 (1.740)
  Change at Week 16: number analyzed (Participants) | 22 | 23 | 19 | 24 | 21
  Change at Week 16 | -1.75 (1.728) | -1.87 (1.915) | -2.39 (2.546) | -1.76 (2.382) | -2.29 (1.630)
  Change at Week 17: number analyzed (Participants) | 19 | 19 | 15 | 20 | 17
  Change at Week 17 | -1.64 (2.182) | -1.85 (1.882) | -2.36 (2.376) | -1.95 (2.282) | -1.97 (1.921)
  Change at Week 18: number analyzed (Participants) | 19 | 20 | 13 | 21 | 16
  Change at Week 18 | -1.47 (2.248) | -2.02 (1.894) | -2.85 (2.521) | -1.95 (2.338) | -1.98 (1.855)
  Change at Week 19: number analyzed (Participants) | 19 | 14 | 15 | 19 | 17
  Change at Week 19 | -1.74 (2.096) | -2.65 (1.508) | -2.93 (2.555) | -1.86 (2.498) | -1.77 (1.756)
  Change at Week 20: number analyzed (Participants) | 17 | 15 | 13 | 18 | 16
  Change at Week 20 | -1.71 (2.207) | -2.51 (1.487) | -2.18 (2.226) | -1.73 (2.575) | -1.96 (1.896)
  Change at Week 21: number analyzed (Participants) | 17 | 14 | 9 | 18 | 13
  Change at Week 21 | -1.98 (2.264) | -2.76 (1.515) | -1.76 (2.227) | -1.99 (2.542) | -1.81 (2.069)
  Change at Week 22: number analyzed (Participants) | 14 | 13 | 11 | 15 | 12
  Change at Week 22 | -1.85 (2.380) | -2.56 (1.833) | -1.75 (2.626) | -1.49 (1.795) | -1.97 (1.941)
  Change at Week 23: number analyzed (Participants) | 16 | 11 | 11 | 12 | 9
  Change at Week 23 | -1.36 (2.701) | -2.12 (2.012) | -1.59 (2.168) | -1.20 (1.647) | -1.59 (2.473)
  Change at Week 24: number analyzed (Participants) | 13 | 10 | 10 | 13 | 10
  Change at Week 24 | -2.00 (2.278) | -2.11 (2.083) | -1.84 (2.290) | -0.94 (1.625) | -1.58 (1.952)

3. Secondary Outcome: Percentage of Participants Who Achieved At Least 30 Percent (%) and 50% Reduction in Mean Average Daily Pain Score
Description: as for outcome 1
Time Frame: Week 8, 16
Population: ITT analysis set included all randomized participants who had received at least 1 dose of study medication. Missing values were imputed using baseline observation carried forward (BOCF) method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
percentage of participants
  Week 8: At least 30% Reduction | 35.7 | 26.8 | 35.1 | 35.0 | 35.0
  Week 8: At least 50% Reduction | 21.4 | 14.6 | 24.3 | 25.0 | 17.5
  Week 16: At least 30% Reduction | 33.3 | 31.7 | 35.1 | 27.5 | 27.5
  Week 16: At least 50% Reduction | 19.0 | 17.1 | 24.3 | 15.0 | 20.0
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 1 mg; Week 8, at least 30% Reduction: Logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.660, 95% CI 2-sided [0.259 to 1.683]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.975, 95% CI 2-sided [0.387 to 2.457]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.969, 95% CI 2-sided [0.392 to 2.398]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.969, 95% CI 2-sided [0.392 to 2.398]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 1 mg; Week 8, at least 50% Reduction: Logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.629, 95% CI 2-sided [0.202 to 1.960]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 1.179, 95% CI 2-sided [0.411 to 3.376]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 1.222, 95% CI 2-sided [0.438 to 3.414]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; Odds Ratio (OR) = 0.778, 95% CI 2-sided [0.259 to 2.335]
Statistical Analysis 9: Comparison: Placebo vs Tanezumab 1 mg; Week 16, at least 30% Reduction: Logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.929, 95% CI 2-sided [0.370 to 2.327]
Statistical Analysis 10: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; Odds Ratio (OR) = 1.083, 95% CI 2-sided [0.427 to 2.749]
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; Odds Ratio (OR) = 0.759, 95% CI 2-sided [0.295 to 1.952]
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; Odds Ratio (OR) = 0.759, 95% CI 2-sided [0.295 to 1.952]
Statistical Analysis 13: Comparison: Placebo vs Tanezumab 1 mg; Week 16, at least 50% Reduction: Logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.875, 95% CI 2-sided [0.285 to 2.682]
Statistical Analysis 14: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; Odds Ratio (OR) = 1.366, 95% CI 2-sided [0.466 to 4.006]
Statistical Analysis 15: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; Odds Ratio (OR) = 0.750, 95% CI 2-sided [0.235 to 2.394]
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; Odds Ratio (OR) = 1.063, 95% CI 2-sided [0.356 to 3.168]

4. Secondary Outcome: Change From Baseline in Mean Worst Daily Pain Score at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24
Description: Worst daily pain score was defined as the mean of the last 7 daily diary pain ratings prior to each assessment time point. Participants rated their worst bladder pain due to IC/PBS over the past 24 hours on an 11-point NRS ranging from 0 = no bladder pain to 10 = worst possible bladder pain.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
units on a scale
  Baseline | 6.84 (1.341) | 7.29 (1.489) | 7.32 (1.263) | 7.15 (1.342) | 7.41 (1.334)
  Change at Week 1: number analyzed (Participants) | 42 | 41 | 36 | 39 | 40
  Change at Week 1 | -0.37 (1.097) | -0.45 (1.038) | -0.76 (1.797) | -0.33 (0.966) | -0.49 (0.954)
  Change at Week 2: number analyzed (Participants) | 41 | 41 | 36 | 39 | 40
  Change at Week 2 | -0.84 (1.363) | -0.60 (1.212) | -0.98 (2.078) | -0.72 (1.582) | -0.98 (1.230)
  Change at Week 3: number analyzed (Participants) | 41 | 39 | 35 | 39 | 39
  Change at Week 3 | -0.96 (1.590) | -0.80 (1.785) | -1.03 (1.970) | -1.07 (1.788) | -1.11 (1.290)
  Change at Week 4: number analyzed (Participants) | 40 | 36 | 34 | 37 | 39
  Change at Week 4 | -0.87 (1.660) | -1.12 (1.967) | -1.36 (2.083) | -1.52 (2.074) | -1.42 (1.853)
  Change at Week 5: number analyzed (Participants) | 39 | 36 | 31 | 36 | 37
  Change at Week 5 | -1.00 (1.859) | -1.13 (1.712) | -1.31 (2.215) | -1.71 (2.306) | -1.69 (1.505)
  Change at Week 6: number analyzed (Participants) | 38 | 35 | 30 | 35 | 36
  Change at Week 6 | -0.85 (1.784) | -1.50 (1.953) | -1.53 (2.321) | -1.48 (2.248) | -1.53 (1.715)
  Change at Week 7: number analyzed (Participants) | 40 | 31 | 30 | 34 | 36
  Change at Week 7 | -1.06 (1.963) | -1.59 (2.163) | -1.45 (2.297) | -1.77 (2.324) | -1.73 (1.958)
  Change at Week 8: number analyzed (Participants) | 38 | 32 | 31 | 34 | 34
  Change at Week 8 | -1.20 (1.927) | -1.07 (1.831) | -1.30 (2.462) | -1.68 (2.415) | -1.78 (1.751)
  Change at Week 9: number analyzed (Participants) | 37 | 29 | 28 | 31 | 31
  Change at Week 9 | -1.18 (1.940) | -1.32 (2.227) | -1.51 (2.401) | -1.74 (2.501) | -1.92 (1.679)
  Change at Week 10: number analyzed (Participants) | 33 | 26 | 25 | 28 | 30
  Change at Week 10 | -1.30 (2.050) | -1.02 (2.078) | -1.95 (2.449) | -1.77 (2.181) | -2.13 (2.000)
  Change at Week 11: number analyzed (Participants) | 32 | 28 | 23 | 29 | 29
  Change at Week 11 | -1.41 (1.999) | -1.31 (2.185) | -1.92 (2.334) | -2.00 (2.677) | -2.19 (2.209)
  Change at Week 12: number analyzed (Participants) | 31 | 27 | 24 | 28 | 29
  Change at Week 12 | -1.56 (1.836) | -1.06 (2.075) | -1.73 (2.175) | -1.84 (2.787) | -2.06 (2.056)
  Change at Week 13: number analyzed (Participants) | 33 | 26 | 23 | 25 | 29
  Change at Week 13 | -1.49 (1.937) | -1.20 (2.109) | -1.82 (2.250) | -1.86 (2.617) | -2.35 (2.098)
  Change at Week 14: number analyzed (Participants) | 32 | 24 | 23 | 24 | 27
  Change at Week 14 | -1.49 (1.982) | -1.15 (2.319) | -1.54 (1.903) | -1.69 (2.611) | -2.00 (2.116)
  Change at Week 15: number analyzed (Participants) | 28 | 24 | 22 | 25 | 23
  Change at Week 15 | -1.34 (1.858) | -1.40 (2.138) | -1.64 (1.881) | -1.80 (2.608) | -2.12 (2.212)
  Change at Week 16: number analyzed (Participants) | 22 | 23 | 19 | 24 | 21
  Change at Week 16 | -1.66 (1.878) | -1.48 (2.317) | -2.21 (2.405) | -1.89 (2.547) | -2.39 (2.107)
  Change at Week 17: number analyzed (Participants) | 19 | 19 | 15 | 20 | 17
  Change at Week 17 | -1.48 (2.138) | -1.27 (2.339) | -1.83 (2.228) | -1.93 (2.568) | -2.08 (2.273)
  Change at Week 18: number analyzed (Participants) | 19 | 20 | 13 | 21 | 16
  Change at Week 18 | -1.34 (2.066) | -1.50 (2.275) | -2.53 (2.530) | -2.06 (2.761) | -1.99 (2.105)
  Change at Week 19: number analyzed (Participants) | 19 | 14 | 15 | 19 | 17
  Change at Week 19 | -1.54 (2.388) | -1.92 (2.827) | -2.68 (2.717) | -1.92 (2.916) | -1.66 (2.184)
  Change at Week 20: number analyzed (Participants) | 17 | 15 | 13 | 18 | 16
  Change at Week 20 | -1.42 (2.318) | -1.56 (2.517) | -1.79 (2.393) | -1.85 (2.990) | -1.85 (2.068)
  Change at Week 21: number analyzed (Participants) | 17 | 14 | 9 | 18 | 13
  Change at Week 21 | -1.73 (2.356) | -1.81 (2.344) | -1.35 (1.695) | -2.24 (2.975) | -1.64 (2.246)
  Change at Week 22: number analyzed (Participants) | 14 | 13 | 11 | 15 | 12
  Change at Week 22 | -1.69 (2.674) | -1.54 (2.607) | -1.46 (2.425) | -1.62 (2.268) | -1.82 (2.103)
  Change at Week 23: number analyzed (Participants) | 16 | 11 | 11 | 12 | 9
  Change at Week 23 | -1.32 (2.749) | -1.01 (2.686) | -1.45 (1.887) | -1.20 (1.821) | -1.28 (2.562)
  Change at Week 24: number analyzed (Participants) | 13 | 10 | 10 | 13 | 10
  Change at Week 24 | -1.91 (2.701) | -0.80 (2.695) | -1.90 (2.225) | -0.93 (1.738) | -1.48 (2.041)

5. Secondary Outcome: Patient Global Assessment of Health Status Scores
Description: Participants answered: "Considering all the ways your bladder condition (IC/PBS) affects you, how are you doing today?" Participants responded on a 5-point scale where 1 = very good and 5 = very poor.
Time Frame: Baseline, Week 2, 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 35 | 40 | 40
units on a scale
  Baseline | 3.1 (0.58) | 3.1 (0.66) | 3.5 (0.82) | 3.1 (0.61) | 3.1 (0.76)
  Week 2: number analyzed (Participants) | 42 | 41 | 35 | 40 | 38
  Week 2 | 2.7 (0.79) | 2.9 (0.75) | 2.9 (0.90) | 3.0 (0.77) | 2.9 (0.66)
  Week 8: number analyzed (Participants) | 38 | 37 | 28 | 32 | 34
  Week 8 | 2.9 (0.70) | 2.9 (0.94) | 2.9 (0.93) | 2.9 (0.83) | 2.9 (0.90)
  Week 16: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16 | 2.7 (0.73) | 3.0 (0.82) | 2.8 (0.58) | 2.7 (0.88) | 2.8 (0.80)
  Week 24: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24 | 2.7 (0.89) | 2.6 (0.62) | 2.5 (0.94) | 2.8 (0.79) | 3.4 (0.86)

6. Secondary Outcome: Number of Participants With Global Response Assessment Scores
Description: Participants were asked: "compared to when you began this trial, how would you rate your IC/PBS symptoms now?" Participants responded by using a 7-point symmetric scale where 1 = markedly worse, 2 = moderately worse, 3 = slightly worse, 4 = no change, 5 = slightly improved, 6 = moderately improved, and 7 = markedly improved.
Time Frame: Week 8, 16, 24
Population: ITT analysis set. Missing values were imputed using last observation carried forward (LOCF) method. Here 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 38 | 37 | 28 | 33 | 34
Participants
  Week 8: Markedly Worse | 1 | 0 | 1 | 0 | 1
  Week 8: Moderately Worse | 4 | 1 | 2 | 2 | 0
  Week 8: Slightly Worse | 1 | 2 | 1 | 3 | 0
  Week 8: No Change | 13 | 13 | 7 | 11 | 14
  Week 8: Slightly Improved | 8 | 12 | 6 | 9 | 11
  Week 8: Moderately Improved | 8 | 5 | 6 | 4 | 4
  Week 8: Markedly Improved | 3 | 4 | 5 | 4 | 4
  Week 16: Markedly Worse: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Markedly Worse | 1 | 2 | 0 | 1 | 0
  Week 16: Moderately Worse: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Moderately Worse | 3 | 1 | 0 | 0 | 1
  Week 16: Slightly Worse: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Slightly Worse | 1 | 1 | 2 | 2 | 2
  Week 16: No Change: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: No Change | 9 | 12 | 8 | 9 | 13
  Week 16: Slightly Improved: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Slightly Improved | 10 | 8 | 6 | 5 | 8
  Week 16: Moderately Improved: number analyzed (Participants) | 33 | 29 | 23 | 26 | 2
  Week 16: Moderately Improved | 3 | 2 | 5 | 4 | 2
  Week 16: Markedly Improved: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Markedly Improved | 6 | 3 | 2 | 5 | 3
  Week 24: Markedly Worse: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: Markedly Worse | 1 | 0 | 1 | 2 | 0
  Week 24: Moderately Worse: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: Moderately Worse | 0 | 3 | 1 | 2 | 1
  Week 24: Slightly Worse: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: Slightly Worse | 2 | 1 | 1 | 2 | 0
  Week 24: No Change: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: No Change | 7 | 4 | 7 | 4 | 5
  Week 24: Slightly Improved: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: Slightly Improved | 4 | 5 | 3 | 4 | 5
  Week 24: Moderately Improved: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: Moderately Improved | 3 | 3 | 1 | 3 | 4
  Week 24: Markedly Improved: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Week 24: Markedly Improved | 2 | 1 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 1 mg; Week 8: Proportional odds logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; p = 0.5731, Regression, Logistic; Odds Ratio (OR) = 1.263, 95% CI 2-sided [0.560 to 2.848]
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 2.5 mg; Week 8: Proportional odds logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; p = 0.2592, Regression, Logistic; Odds Ratio (OR) = 1.656, 95% CI 2-sided [0.689 to 3.980]
Statistical Analysis 3: Comparison: Placebo vs Tanezumab 10 mg; Week 8: Proportional odds logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; p = 1.045, Regression, Logistic; Odds Ratio (OR) = 0.9181, 95% CI 2-sided [0.452 to 2.417]
Statistical Analysis 4: Comparison: Placebo vs Tanezumab 20 mg; Week 8: Proportional odds logistic regression analysis with treatment as independent variable was used for the analysis; Test type: Superiority or Other; p = 0.5289, Regression, Logistic; Odds Ratio (OR) = 1.306, 95% CI 2-sided [0.569 to 2.997]
Statistical Analysis 5: Comparison: Placebo vs Tanezumab 1 mg; Week 16: Proportional odds logistic regression analysis with treatment as independent variable was used for the analysis. For Week 16, data scores were combined into 3 categories: Improved ('slightly improved', 'moderately improved', 'markedly improved'), No Change ('no change') and Worse ('markedly worse', 'moderately worse', 'slightly worse') for comparison; Test type: Superiority or Other; p = 0.7930, Regression, Logistic; Odds Ratio (OR) = 0.893, 95% CI 2-sided [0.385 to 2.074]
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 2.5 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.7386, Regression, Logistic; Odds Ratio (OR) = 1.167, 95% CI 2-sided [0.471 to 2.892]
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.9354, Regression, Logistic; Odds Ratio (OR) = 1.036, 95% CI 2-sided [0.437 to 2.460]
Statistical Analysis 8: Comparison: Placebo vs Tanezumab 20 mg; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.6207, Regression, Logistic; Odds Ratio (OR) = 0.805, 95% CI 2-sided [0.341 to 1.899]

7. Secondary Outcome: Number of Micturitions Per 24 Hours
Description: The micturition frequency per 24 hours was calculated from the sum of voids divided by the diary period over which they were collected.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 41 | 39 | 37 | 40 | 40
micturitions per 24 hours
  Baseline | 12.98 (5.207) | 13.04 (5.500) | 14.12 (6.728) | 13.27 (5.403) | 13.13 (5.681)
  Week 4: number analyzed (Participants) | 31 | 34 | 29 | 26 | 30
  Week 4 | 11.03 (4.867) | 11.81 (6.843) | 11.41 (5.735) | 10.62 (6.635) | 13.14 (7.930)
  Week 8: number analyzed (Participants) | 30 | 30 | 30 | 30 | 31
  Week 8 | 11.61 (5.662) | 12.18 (6.675) | 10.39 (4.842) | 11.52 (7.009) | 11.13 (7.754)
  Week 12: number analyzed (Participants) | 21 | 24 | 20 | 19 | 24
  Week 12 | 10.19 (5.265) | 12.88 (7.234) | 10.58 (4.933) | 10.21 (6.185) | 10.15 (5.695)
  Week 16: number analyzed (Participants) | 20 | 23 | 17 | 22 | 18
  Week 16 | 9.24 (4.940) | 11.27 (4.892) | 10.93 (3.810) | 8.90 (6.212) | 9.99 (5.355)
  Week 20: number analyzed (Participants) | 12 | 15 | 14 | 15 | 14
  Week 20 | 10.82 (6.034) | 12.11 (5.985) | 9.61 (4.987) | 10.17 (7.354) | 12.26 (7.272)
  Week 24: number analyzed (Participants) | 10 | 10 | 10 | 11 | 9
  Week 24 | 11.10 (6.190) | 10.67 (5.871) | 10.67 (5.571) | 11.36 (5.575) | 11.04 (6.417)

8. Secondary Outcome: Number of Nocturnal Micturitions Per 24 Hours
Description: The nocturnal frequency per 24 hours was defined as the number of voids after going to bed and before getting up (the times of going to bed and getting up were recorded in the diary). The nocturnal micturition per 24 hours was calculated as the sum of voluntary voids that occurred during a night's sleep, divided by the number of nights over which this was collected.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 41 | 40 | 37 | 40 | 40
micturitions per 24 hours
  Baseline | 2.63 (1.641) | 3.34 (2.379) | 2.66 (1.850) | 3.39 (2.667) | 2.95 (1.761)
  Week 4: number analyzed (Participants) | 31 | 34 | 29 | 27 | 31
  Week 4 | 2.25 (1.634) | 3.40 (2.904) | 2.85 (1.720) | 2.44 (2.671) | 2.72 (2.601)
  Week 8: number analyzed (Participants) | 30 | 30 | 30 | 30 | 32
  Week 8 | 2.58 (1.982) | 3.18 (2.094) | 2.44 (1.851) | 3.12 (3.316) | 2.73 (2.258)
  Week 12: number analyzed (Participants) | 23 | 25 | 20 | 21 | 25
  Week 12 | 1.97 (1.326) | 2.87 (2.023) | 2.62 (1.371) | 2.02 (2.106) | 2.71 (2.023)
  Week 16: number analyzed (Participants) | 20 | 23 | 18 | 23 | 20
  Week 16 | 2.45 (3.141) | 3.55 (2.982) | 2.77 (1.456) | 2.17 (1.789) | 2.31 (1.949)
  Week 20: number analyzed (Participants) | 13 | 16 | 13 | 16 | 14
  Week 20 | 2.95 (3.031) | 4.60 (4.302) | 2.29 (1.279) | 2.96 (2.937) | 3.89 (3.129)
  Week 24: number analyzed (Participants) | 12 | 10 | 10 | 12 | 9
  Week 24 | 2.15 (1.693) | 3.45 (2.132) | 2.68 (1.426) | 3.39 (3.731) | 2.56 (1.891)

9. Secondary Outcome: Number of Micturition-related Urgency Episodes Per 24 Hours
Description: The micturition urgency frequency per 24 hours was calculated as the sum of urgency episodes (when participant had to rush to get to the bathroom to urinate) occurring during the diary period when this was measured, divided by the number of days over which they were recorded.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: urgency episodes per 24 hours
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 41 | 39 | 37 | 40 | 40
urgency episodes per 24 hours
  Baseline | 6.88 (6.721) | 7.04 (6.040) | 9.24 (7.665) | 8.38 (5.774) | 7.20 (6.842)
  Week 4: number analyzed (Participants) | 31 | 34 | 28 | 26 | 30
  Week 4 | 4.64 (5.680) | 6.90 (7.560) | 8.27 (10.391) | 5.97 (4.849) | 6.91 (8.820)
  Week 8: number analyzed (Participants) | 29 | 30 | 30 | 30 | 31
  Week 8 | 6.06 (7.493) | 6.50 (7.674) | 5.86 (5.213) | 6.51 (7.504) | 6.23 (8.625)
  Week 12: number analyzed (Participants) | 21 | 24 | 20 | 19 | 24
  Week 12 | 4.90 (6.575) | 5.73 (5.419) | 5.89 (5.035) | 5.09 (4.852) | 5.31 (6.597)
  Week 16: number analyzed (Participants) | 19 | 23 | 17 | 22 | 18
  Week 16 | 4.78 (6.254) | 5.06 (4.473) | 6.52 (6.374) | 4.34 (4.940) | 6.01 (6.511)
  Week 20: number analyzed (Participants) | 12 | 15 | 14 | 15 | 14
  Week 20 | 3.81 (5.482) | 4.62 (5.341) | 5.37 (5.840) | 5.09 (5.565) | 7.40 (8.167)
  Week 24: number analyzed (Participants) | 10 | 10 | 10 | 10 | 9
  Week 24 | 4.53 (6.286) | 3.65 (5.695) | 6.80 (6.568) | 6.62 (8.546) | 6.43 (7.734)

10. Secondary Outcome: Participant's Urge to Urinate
Description: Participants completed 7-item questionnaire assessing their urge to urinate over the past 24 hours. The items were assessed on a 5-point response scale ranging from 0 (never) to 4 (always). Urge to urinate was calculated as the total of the 7 'urge' items with a minimum total score of 0 and a maximum total score of 28. Higher scores indicated greater symptom severity. An average was determined from the 3 days recorded in the 7-day diary period prior to each assessment time point.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
units on a scale
  Baseline | 15.63 (4.313) | 17.04 (5.015) | 18.95 (4.750) | 17.73 (3.794) | 17.11 (5.011)
  Week 4: number analyzed (Participants) | 34 | 36 | 31 | 28 | 31
  Week 4 | 13.75 (5.871) | 16.27 (5.990) | 14.87 (5.750) | 15.71 (4.699) | 14.83 (6.234)
  Week 8: number analyzed (Participants) | 31 | 31 | 30 | 31 | 31
  Week 8 | 14.81 (4.951) | 15.80 (6.338) | 14.71 (6.297) | 14.38 (4.804) | 13.81 (6.830)
  Week 12: number analyzed (Participants) | 24 | 26 | 20 | 23 | 29
  Week 12 | 13.21 (6.010) | 15.64 (6.904) | 13.75 (6.376) | 14.43 (5.635) | 14.02 (7.761)
  Week 16: number analyzed (Participants) | 20 | 23 | 18 | 24 | 22
  Week 16 | 13.59 (5.589) | 14.28 (6.083) | 13.49 (6.223) | 14.05 (5.812) | 13.85 (8.156)
  Week 20: number analyzed (Participants) | 14 | 16 | 14 | 19 | 14
  Week 20 | 14.05 (5.729) | 12.75 (7.124) | 11.95 (7.226) | 13.97 (5.887) | 15.62 (9.020)
  Week 24: number analyzed (Participants) | 12 | 12 | 10 | 13 | 10
  Week 24 | 12.39 (7.258) | 13.25 (6.489) | 11.13 (7.442) | 14.28 (4.870) | 15.87 (8.800)

11. Secondary Outcome: Mean Voided Volume Per Micturition
Description: Mean volume voided per micturition was calculated as the total urine volume voided during the diary period when this was measured over 1 day, divided by the number of voids (with non missing volumes) during that day.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 41 | 38 | 37 | 40 | 39
milliliter
  Baseline | 142.12 (68.374) | 129.58 (57.649) | 122.78 (65.259) | 146.71 (71.013) | 139.92 (71.064)
  Week 4: number analyzed (Participants) | 31 | 32 | 27 | 25 | 29
  Week 4 | 130.75 (57.303) | 144.48 (110.219) | 117.45 (59.046) | 175.99 (97.418) | 140.84 (91.375)
  Week 8: number analyzed (Participants) | 29 | 29 | 28 | 29 | 30
  Week 8 | 132.33 (57.848) | 148.56 (109.210) | 165.02 (114.862) | 152.77 (86.116) | 155.09 (106.398)
  Week 12: number analyzed (Participants) | 21 | 22 | 19 | 20 | 22
  Week 12 | 136.60 (64.056) | 164.68 (180.771) | 136.06 (88.539) | 180.01 (85.147) | 158.35 (119.294)
  Week 16: number analyzed (Participants) | 19 | 23 | 16 | 21 | 19
  Week 16 | 141.39 (67.788) | 117.78 (75.291) | 112.86 (66.617) | 180.71 (88.065) | 163.20 (128.409)
  Week 20: number analyzed (Participants) | 13 | 16 | 12 | 14 | 12
  Week 20 | 131.52 (61.604) | 118.44 (68.203) | 139.61 (64.196) | 189.66 (86.580) | 135.80 (95.869)
  Week 24: number analyzed (Participants) | 10 | 10 | 10 | 10 | 9
  Week 24 | 138.77 (87.222) | 124.48 (76.990) | 152.99 (102.429) | 182.66 (95.542) | 174.96 (118.350)

12. Secondary Outcome: O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) Score
Description: The ICSI contained 4 questions that measured symptom severity including urinary urgency, urinary frequency, nocturia and pain/burning in the bladder. Each question in the ICSI was rated on a 0-5 scale. The sum of the individual question ratings was the total score for the ICSI. Total scores ranged from 0 to 20, with higher scores indicating greater symptom severity and bother.
Time Frame: Baseline, Week 2, 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 36 | 40 | 39
units on a scale
  Baseline: number analyzed (Participants) | 42 | 41 | 35 | 40 | 39
  Baseline | 13.1 (3.39) | 14.1 (3.15) | 15.2 (3.25) | 14.4 (2.78) | 14.5 (2.72)
  Week 2: number analyzed (Participants) | 42 | 41 | 36 | 40 | 38
  Week 2 | 11.2 (3.74) | 13.1 (3.72) | 13.2 (4.62) | 12.9 (3.66) | 13.0 (3.82)
  Week 8: number analyzed (Participants) | 38 | 37 | 28 | 33 | 34
  Week 8 | 11.4 (3.26) | 12.7 (4.44) | 12.6 (5.06) | 12.2 (4.23) | 12.2 (4.70)
  Week 16: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16 | 10.8 (4.22) | 13.4 (3.77) | 12.5 (4.47) | 11.5 (4.89) | 12.3 (4.92)
  Week 24: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24 | 11.9 (4.79) | 12.3 (5.06) | 12.2 (4.67) | 12.2 (4.33) | 11.5 (5.61)

13. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-sf) Score
Description: BPI-sf is a 7-item self-administered questionnaire to assess the pain severity and pain interference on daily functions. Pain Severity Index (PSI) is an average of Questions 2-5 which measured the severity of pain (worst, least, average, right now) over past 24-hours on an 11-point scale (0=no pain to 10=pain as bad as you can imagine). Pain Interference Index (PII) is an average of 7 pain interference items of Question 7 that measured the level of interference of pain on daily function (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life) on an 11-point scale (0=did not interfere to 10=completely interfered). Pain Severity Index and Pain Interference Index total scores ranged from 0 to 10, where higher scores indicate greater pain or greater interference.
Time Frame: Baseline, Week 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 35 | 40 | 40
units on a scale
  Baseline: PSI | 5.14 (1.387) | 5.28 (1.788) | 5.74 (1.817) | 5.49 (1.904) | 5.82 (1.491)
  Baseline: PII | 4.80 (1.963) | 5.22 (2.082) | 5.49 (2.251) | 4.97 (1.932) | 5.74 (1.808)
  Week 8: PSI: number analyzed (Participants) | 38 | 37 | 28 | 33 | 34
  Week 8: PSI | 4.12 (2.072) | 4.28 (2.090) | 4.84 (2.318) | 4.30 (2.293) | 4.60 (1.984)
  Week 8: PII: number analyzed (Participants) | 38 | 37 | 28 | 33 | 34
  Week 8: PII | 3.76 (2.432) | 4.49 (2.607) | 4.46 (2.980) | 3.93 (2.513) | 4.61 (2.598)
  Week 16: PSI: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: PSI | 3.86 (2.023) | 4.53 (2.238) | 4.21 (2.136) | 4.23 (2.417) | 4.51 (1.912)
  Week 16: PII: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: PII | 3.59 (2.511) | 4.67 (2.552) | 4.52 (2.715) | 3.87 (2.600) | 4.31 (2.467)
  Week 24: PSI: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: PSI | 3.96 (2.159) | 3.16 (1.871) | 3.99 (2.376) | 4.57 (2.001) | 5.16 (1.879)
  Week 24, PII: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24, PII | 4.16 (2.153) | 3.53 (2.739) | 4.48 (3.149) | 4.54 (2.246) | 4.39 (2.699)

14. Secondary Outcome: Number of Participants With Patient Global Satisfaction Assessment Scores
Description: Participant global satisfaction is assessed using Patient Reported Treatment Impact (PRTI) which is a self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participants were asked: "Overall, how satisfied are you with the drug that you received since you entered this trial?" Participant's response is rated on a 5-point scale where 1=extremely dissatisfied (dissatisf), 2=dissatisfied, 3=neither satisfied nor dissatisfied (satisfy/dissatisfy), 4=satisfied and 5=extremely satisfied. Number of participants with each response is reported.
Time Frame: Week 8, 16, 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 38 | 36 | 28 | 32 | 34
Participants
  Week 8: Extremely Satisfied | 5 | 3 | 7 | 5 | 5
  Week 8: Satisfied | 12 | 11 | 8 | 5 | 9
  Week 8: Satisfy/Dissatisfy | 14 | 14 | 6 | 17 | 11
  Week 8: Dissatisfied | 6 | 4 | 7 | 3 | 5
  Week 8: Extremely Dissatisf | 1 | 4 | 0 | 2 | 4
  Week 16: Extremely Satisfied: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Extremely Satisfied | 3 | 6 | 4 | 5 | 3
  Week 16: Satisfied: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Satisfied | 12 | 5 | 7 | 5 | 5
  Week16: Satisfy/Dissatisfy: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week16: Satisfy/Dissatisfy | 11 | 10 | 8 | 11 | 12
  Week 16: Dissatisfied: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Dissatisfied | 6 | 7 | 3 | 1 | 4
  Week 16: Extremely Dissatisf: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Extremely Dissatisf | 1 | 1 | 1 | 4 | 5
  Week 24: Extremely Satisfied: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Extremely Satisfied | 6 | 4 | 6 | 5 | 4
  Week 24: Satisfied: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Satisfied | 4 | 5 | 2 | 5 | 5
  Week 24: Satisfy/Dissatisfy: number analyzed (Participants) | 19 | 17 | 17 | 8 | 17
  Week 24: Satisfy/Dissatisfy | 7 | 3 | 7 | 5 | 6
  Week 24: Dissatisfied: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Dissatisfied | 1 | 1 | 1 | 0 | 0
  Week 24: Extremely Dissatisf: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Extremely Dissatisf | 1 | 4 | 1 | 3 | 2

15. Secondary Outcome: Number of Participants With Patient Global Preference Assessment Score
Description: Participant global preference is assessed using PRTI which is self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment (T/T), preference and willingness to continue using study medication. Participant reported previous T/T under following categories: lifestyle interventions, physical therapies, toileting programs, drug given into bladder, drug taken by mouth, surgery, and no T/T. Participant preference was assessed on a 5-point scale where, 1=No, I definitely prefer my prior T/T (Def Pref Prior), 2=I have a slight preference for my prior T/T (Slight Pref Prior T/T), 3=I have no preference either way (No preference), 4=I have a slight preference for the drug that I am receiving now (Slight Pref Current), 5=Yes, I definitely prefer the drug that I am receiving (Def Pref Current Drug) now. Number of participants under each of the categories is reported. For previous T/T, a single participant may be represented in more than 1 category.
Time Frame: Week 8, 16, 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 38 | 36 | 28 | 32 | 34
Participants
  Week 8: Lifestyle Interventions | 16 | 17 | 16 | 17 | 14
  Week 8: Physical Therapies | 8 | 4 | 5 | 8 | 6
  Week 8: Toileting Programs | 2 | 1 | 1 | 0 | 1
  Week 8: Drug Given Into Bladder | 7 | 9 | 9 | 8 | 11
  Week 8: Drug Taken by Mouth | 24 | 20 | 17 | 22 | 20
  Week 8: Surgery | 3 | 3 | 5 | 4 | 6
  Week 8: No Treatment | 6 | 2 | 4 | 3 | 4
  Week 8: Def Pref Current Drug | 9 | 11 | 7 | 7 | 7
  Week 8:Slight Pref Current | 9 | 8 | 8 | 6 | 10
  Week 8: No Preference | 14 | 12 | 8 | 15 | 10
  Week8:Slight Pref Prior T/T | 4 | 2 | 2 | 2 | 3
  Week 8: Def Pref Prior | 2 | 3 | 3 | 2 | 4
  Week 16:Lifestyle Interventions: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16:Lifestyle Interventions | 15 | 14 | 9 | 12 | 12
  Week 16: Physical Therapies: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Physical Therapies | 6 | 4 | 4 | 5 | 8
  Week 16: Toileting Programs: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16: Toileting Programs | 2 | 2 | 4 | 0 | 2
  Week 16:Drug Given Into Bladder: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16:Drug Given Into Bladder | 5 | 8 | 9 | 4 | 9
  Week 16: Drug Taken by Mouth: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16: Drug Taken by Mouth | 21 | 17 | 11 | 16 | 16
  Week 16: Surgery: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16: Surgery | 5 | 3 | 3 | 3 | 4
  Week 16: No Treatment: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16: No Treatment | 6 | 2 | 6 | 3 | 4
  Week 16: Def Pref Current Drug: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16: Def Pref Current Drug | 8 | 8 | 6 | 7 | 5
  Week 16:Slight Pref Current: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16:Slight Pref Current | 7 | 8 | 7 | 8 | 8
  Week 16: No Preference: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16: No Preference | 16 | 7 | 8 | 9 | 10
  Week16:Slight Pref Prior T/T: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week16:Slight Pref Prior T/T | 1 | 4 | 1 | 0 | 1
  Week 16:Def Pref Prior: number analyzed (Participants) | 38 | 29 | 23 | 26 | 29
  Week 16:Def Pref Prior | 1 | 2 | 1 | 2 | 5
  Week 24:Lifestyle Interventions: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24:Lifestyle Interventions | 8 | 7 | 10 | 7 | 7
  Week 24: Physical Therapies: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Physical Therapies | 6 | 2 | 4 | 6 | 7
  Week 24: Toileting Programs: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Toileting Programs | 2 | 1 | 2 | 0 | 0
  Week 24:Drug Given Into Bladder: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24:Drug Given Into Bladder | 3 | 4 | 9 | 6 | 6
  Week 24: Drug Taken by Mouth: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Drug Taken by Mouth | 12 | 9 | 12 | 12 | 11
  Week 24: Surgery: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Surgery | 1 | 3 | 4 | 4 | 4
  Week 24: No Treatment: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: No Treatment | 2 | 2 | 1 | 1 | 1
  Week 24: Def Pref Current Drug: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Def Pref Current Drug | 6 | 4 | 6 | 5 | 4
  Week 24:Slight Pref Current: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24:Slight Pref Current | 4 | 5 | 2 | 5 | 5
  Week 24: No Preference: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: No Preference | 7 | 3 | 7 | 5 | 6
  Week 24: Slight Pref Prior T/T: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Slight Pref Prior T/T | 1 | 1 | 1 | 0 | 0
  Week 24:Def Pref Prior: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24:Def Pref Prior | 1 | 4 | 1 | 3 | 2

16. Secondary Outcome: Number of Participants With Willingness to Re-use Medicine Assessment
Description: Participant willingness to re-use study medication is assessed using PRTI which is a self-administered questionnaire containing four items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. Participants were asked: "In the future, would you be willing to use the same drug that you have received since you entered this trial for your chronic prostatitis?" Participants responded on 5-point scale where, 1=No, I definitely would not want to use the same drug again (definitely not want), 2=I might not want to use the same drug again (might not want), 3=I am not sure (not sure), 4=I might want to use the same drug again (might want), 5=Yes, I would definitely want to use the same drug again (definitely want).
Time Frame: Week 8, 16, 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 38 | 36 | 28 | 32 | 33
Participants
  Week 8: Definitely Want | 12 | 12 | 10 | 10 | 12
  Week 8: Might Want | 11 | 10 | 7 | 9 | 6
  Week 8: Not Sure | 13 | 11 | 7 | 10 | 12
  Week 8: Might not Want | 1 | 0 | 3 | 1 | 0
  Week 8: Definitely not Want | 1 | 3 | 1 | 2 | 3
  Week 16: Definitely Want: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Definitely Want | 3 | 6 | 4 | 5 | 3
  Week 16: Might Want: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Might Want | 12 | 5 | 7 | 5 | 5
  Week 16: Not Sure: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Not Sure | 11 | 10 | 8 | 11 | 12
  Week 16: Might not Want: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Might not Want | 6 | 7 | 3 | 1 | 4
  Week 16: Definitely not Want: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16: Definitely not Want | 1 | 1 | 1 | 4 | 5
  Week 24: Definitely Want: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Definitely Want | 6 | 5 | 7 | 7 | 6
  Week 24: Might Want: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Might Want | 4 | 2 | 4 | 2 | 0
  Week 24: Not Sure: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Not Sure | 4 | 7 | 5 | 6 | 5
  Week 24: Might not Want: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Might not Want | 3 | 1 | 1 | 0 | 2
  Week 24: Definitely not Want: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24: Definitely not Want | 2 | 2 | 0 | 3 | 4

17. Secondary Outcome: Euro Quality of Life (EQ-5D) - Health State Profile Utility Score
Description: EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Week 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 35 | 40 | 39
units on a scale
  Baseline | 0.69 (0.209) | 0.68 (0.182) | 0.56 (0.233) | 0.70 (0.167) | 0.61 (0.224)
  Week 8: number analyzed (Participants) | 38 | 37 | 28 | 32 | 34
  Week 8 | 0.74 (0.235) | 0.73 (0.191) | 0.69 (0.214) | 0.70 (0.185) | 0.68 (0.233)
  Week 16: number analyzed (Participants) | 33 | 29 | 23 | 26 | 29
  Week 16 | 0.75 (0.221) | 0.71 (0.187) | 0.72 (0.162) | 0.77 (0.124) | 0.73 (0.215)
  Week 24: number analyzed (Participants) | 19 | 17 | 17 | 18 | 17
  Week 24 | 0.74 (0.174) | 0.76 (0.187) | 0.72 (0.232) | 0.67 (0.202) | 0.66 (0.252)

18. Secondary Outcome: Painful Bladder/Interstitial Cystitis Quality of Life Questionnaire (PBIC-QoL) Total Score
Description: PBIC-QoL: 25-item questionnaire to assess impact of IC/PBS on health related quality of life over past 7 days. PBIC-QoL included 17 items (Items 2, 5, 8, 11, 14, 18, 20 and 21 did not form part of final instrument), of which 13 were divided into 3 dimensions: activity limitations (Items 1, 3, 4, 6, 7), impact on emotional wellbeing (Items 13, 15, 16, 17, 19), impact on sleep (Items 22, 23, 24). Four items: Item 9 (impact on going out with friends), Item 10 (impact on concentration), Item 12 (impact on eating and drinking), Item 25 (impact on sex life) were scored separately to dimension scores as single items. Items were scored from 4 'not at all' to 0 'extremely difficult' or 'a very great deal'. Eight items included a 'not applicable' response option. Dimension scores ranged from 0 to 4, higher score indicate better quality of life. Total score=sum of the dimension and single item scores, ranged from 0 to 28, higher score indicated better quality of life.
Time Frame: Baseline, Week 2, 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 24 | 31 | 27 | 25 | 30
units on a scale
  Baseline: number analyzed (Participants) | 24 | 31 | 26 | 25 | 30
  Baseline | 11.49 (4.774) | 10.56 (4.147) | 10.39 (5.531) | 11.44 (3.938) | 10.42 (5.172)
  Week 2: number analyzed (Participants) | 22 | 29 | 27 | 25 | 28
  Week 2 | 16.41 (5.784) | 12.79 (5.173) | 13.77 (6.953) | 15.34 (5.895) | 13.24 (6.093)
  Week 8: number analyzed (Participants) | 23 | 24 | 22 | 20 | 25
  Week 8 | 16.47 (5.256) | 12.02 (5.594) | 15.26 (7.272) | 14.42 (6.635) | 14.10 (6.606)
  Week 16: number analyzed (Participants) | 22 | 19 | 17 | 18 | 22
  Week 16 | 16.49 (6.180) | 11.19 (4.486) | 15.21 (6.671) | 17.23 (5.868) | 13.94 (7.153)
  Week 24: number analyzed (Participants) | 13 | 9 | 13 | 12 | 14
  Week 24 | 14.27 (7.808) | 14.45 (5.663) | 16.77 (8.044) | 14.27 (5.813) | 15.05 (6.852)

19. Secondary Outcome: Percentage of Participants Who Received Rescue Medication
Description: For inadequate pain relief or worsening symptoms of IC/PBS, participants took acetaminophen up to 3000 mg per day (1500 mg/day for Japanese population) as rescue medication.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: ITT analysis set included all randomized participants who had received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
percentage of participants
  Baseline | 52.4 | 65.9 | 56.8 | 50.0 | 57.5
  Week 1 | 42.9 | 53.7 | 48.6 | 50.0 | 42.5
  Week 2 | 50.0 | 53.7 | 54.1 | 57.5 | 42.5
  Week 3 | 35.7 | 51.2 | 48.6 | 47.5 | 40.0
  Week 4 | 33.3 | 53.7 | 43.2 | 45.0 | 45.0
  Week 5 | 33.3 | 39.0 | 40.5 | 40.0 | 45.0
  Week 6 | 35.7 | 48.8 | 37.8 | 42.5 | 32.5
  Week 7 | 38.1 | 26.8 | 37.8 | 35.0 | 37.5
  Week 8 | 35.7 | 34.1 | 35.1 | 30.0 | 35.0
  Week 9 | 31.0 | 31.7 | 37.8 | 30.0 | 30.0
  Week 10 | 35.7 | 34.1 | 29.7 | 22.5 | 30.0
  Week 11 | 31.0 | 26.8 | 29.7 | 25.0 | 32.5
  Week 12 | 26.2 | 24.4 | 24.3 | 27.5 | 30.0
  Week 13 | 31.0 | 24.4 | 24.3 | 22.5 | 27.5
  Week 14 | 31.0 | 24.4 | 21.6 | 25.0 | 32.5
  Week 15 | 28.6 | 17.1 | 27.0 | 22.5 | 20.0
  Week 16 | 19.0 | 14.6 | 18.9 | 25.0 | 17.5
  Week 17 | 21.4 | 17.1 | 18.9 | 22.5 | 22.5
  Week 18 | 19.0 | 17.1 | 16.2 | 17.5 | 15.0
  Week 19 | 21.4 | 19.5 | 13.5 | 17.5 | 17.5
  Week 20 | 14.3 | 12.2 | 21.6 | 17.5 | 15.0
  Week 21 | 14.3 | 12.2 | 18.9 | 20.0 | 7.5
  Week 22 | 19.0 | 14.6 | 10.8 | 10.8 | 7.5
  Week 23 | 19.0 | 12.2 | 10.8 | 10.0 | 7.5
  Week 24 | 14.3 | 7.3 | 5.4 | 10.0 | 7.5

20. Secondary Outcome: Number of Days of Rescue Medication Usage Per Week
Description: In case of inadequate pain relief or worsening symptoms of IC/PBS, participants took acetaminophen up to 3000 mg per day (1500 mg/day for Japanese population) as rescue medication.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 22 | 27 | 21 | 23 | 23
days per week
  Baseline: number analyzed (Participants) | 22 | 27 | 21 | 20 | 23
  Baseline | 4.1 (2.18) | 3.6 (2.39) | 3.8 (2.27) | 4.1 (2.36) | 4.6 (2.08)
  Week 1: number analyzed (Participants) | 18 | 22 | 18 | 20 | 17
  Week 1 | 4.5 (2.38) | 4.0 (2.21) | 3.8 (2.32) | 4.6 (2.01) | 4.8 (1.68)
  Week 2: number analyzed (Participants) | 21 | 22 | 20 | 23 | 17
  Week 2 | 3.4 (2.56) | 3.9 (2.25) | 3.6 (2.42) | 3.7 (2.38) | 4.2 (2.31)
  Week 3: number analyzed (Participants) | 15 | 21 | 18 | 19 | 16
  Week 3 | 3.5 (2.50) | 3.5 (2.38) | 3.9 (2.49) | 3.6 (2.27) | 4.3 (2.27)
  Week 4: number analyzed (Participants) | 14 | 22 | 16 | 18 | 18
  Week 4 | 3.3 (2.46) | 3.5 (2.42) | 3.1 (2.35) | 3.7 (2.40) | 3.9 (2.63)
  Week 5: number analyzed (Participants) | 14 | 16 | 15 | 16 | 18
  Week 5 | 3.6 (2.37) | 4.6 (2.19) | 3.9 (2.66) | 3.3 (2.57) | 4.2 (2.53)
  Week 6: number analyzed (Participants) | 15 | 20 | 14 | 17 | 13
  Week 6 | 3.7 (2.32) | 3.3 (2.20) | 3.8 (2.22) | 2.22 (2.33) | 4.5 (2.60)
  Week 7: number analyzed (Participants) | 16 | 11 | 14 | 14 | 15
  Week 7 | 3.7 (2.30) | 5.0 (2.00) | 3.9 (2.37) | 3.5 (2.38) | 4.5 (2.36)
  Week 8: number analyzed (Participants) | 15 | 14 | 13 | 12 | 14
  Week 8 | 4.0 (2.07) | 4.6 (1.91) | 3.8 (2.58) | 3.6 (2.61) | 4.3 (2.05)
  Week 9: number analyzed (Participants) | 13 | 13 | 14 | 12 | 12
  Week 9 | 4.2 (1.74) | 4.6 (1.76) | 4.1 (2.37) | 4.1 (2.43) | 3.8 (2.37)
  Week 10: number analyzed (Participants) | 15 | 14 | 11 | 9 | 12
  Week 10 | 3.1 (1.92) | 3.7 (2.05) | 4.4 (2.46) | 4.2 (2.86) | 4.3 (2.46)
  Week 11: number analyzed (Participants) | 13 | 11 | 11 | 10 | 13
  Week 11 | 4.2 (2.24) | 4.0 (2.41) | 4.2 (2.32) | 3.9 (2.64) | 4.1 (2.60)
  Week 12: number analyzed (Participants) | 11 | 10 | 9 | 11 | 12
  Week 12 | 3.6 (2.01) | 4.6 (1.90) | 5.0 (2.50) | 4.1 (2.43) | 3.8 (2.41)
  Week 13: number analyzed (Participants) | 13 | 10 | 9 | 9 | 11
  Week 13 | 3.2 (2.08) | 4.3 (1.64) | 4.7 (2.83) | 4.8 (2.28) | 4.5 (2.21)
  Week 14: number analyzed (Participants) | 13 | 10 | 8 | 10 | 13
  Week 14 | 3.7 (2.46) | 3.8 (2.25) | 4.6 (2.07) | 4.3 (2.58) | 4.1 (2.36)
  Week 15: number analyzed (Participants) | 12 | 7 | 10 | 9 | 8
  Week 15 | 3.2 (2.17) | 4.0 (2.58) | 3.6 (2.59) | 3.3 (2.40) | 5.0 (2.00)
  Week 16: number analyzed (Participants) | 8 | 6 | 7 | 10 | 7
  Week 16 | 3.5 (1.93) | 4.7 (2.16) | 4.1 (1.95) | 3.9 (2.81) | 4.6 (1.27)
  Week 17: number analyzed (Participants) | 9 | 7 | 7 | 9 | 9
  Week 17 | 3.7 (2.45) | 3.3 (2.29) | 4.4 (2.15) | 3.4 (2.46) | 3.7 (2.18)
  Week 18: number analyzed (Participants) | 8 | 7 | 6 | 7 | 6
  Week 18 | 3.6 (2.00) | 3.3 (1.60) | 4.5 (1.64) | 3.1 (2.67) | 4.7 (2.42)
  Week 19: number analyzed (Participants) | 9 | 8 | 5 | 7 | 7
  Week 19 | 3.9 (2.37) | 2.5 (1.41) | 4.6 (2.51) | 3.7 (2.43) | 3.6 (2.57)
  Week 20: number analyzed (Participants) | 6 | 5 | 8 | 7 | 6
  Week 20 | 4.8 (1.72) | 3.2 (2.59) | 4.0 (2.39) | 3.3 (1.98) | 4.0 (2.37)
  Week 21: number analyzed (Participants) | 6 | 5 | 7 | 8 | 3
  Week 21 | 3.8 (2.40) | 3.4 (2.51) | 2.3 (1.38) | 2.4 (2.13) | 5.7 (1.53)
  Week 22: number analyzed (Participants) | 8 | 6 | 4 | 6 | 3
  Week 22 | 3.4 (1.69) | 3.2 (2.14) | 4.3 (2.75) | 3.2 (2.14) | 4.7 (3.21)
  Week 23: number analyzed (Participants) | 8 | 5 | 4 | 4 | 3
  Week 23 | 4.5 (2.07) | 3.6 (2.30) | 4.3 (2.06) | 2.8 (2.22) | 4.7 (3.21)
  Week 24: number analyzed (Participants) | 6 | 3 | 2 | 4 | 3
  Week 24 | 4.5 (2.51) | 4.0 (2.00) | 7.0 (0.00) | 3.3 (2.87) | 5.7 (2.31)

21. Secondary Outcome: Number of Rescue Medication Doses Used Per Week
Description: as for outcome 20
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: doses per week
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
doses per week
  Baseline: number analyzed (Participants) | 22 | 27 | 21 | 20 | 23
  Baseline | 4.09 (2.18) | 3.56 (2.39) | 3.81 (2.27) | 4.10 (2.36) | 4.61 (2.08)
  Week 1: number analyzed (Participants) | 18 | 22 | 18 | 20 | 17
  Week 1 | 4.50 (2.38) | 4.05 (2.21) | 3.78 (2.32) | 4.55 (2.01) | 4.76 (1.68)
  Week 2: number analyzed (Participants) | 21 | 22 | 20 | 23 | 17
  Week 2 | 3.43 (2.56) | 3.86 (2.25) | 3.55 (2.42) | 3.70 (2.38) | 4.24 (2.31)
  Week 3: number analyzed (Participants) | 15 | 21 | 18 | 19 | 16
  Week 3 | 3.53 (2.50) | 3.48 (2.38) | 3.89 (2.49) | 3.58 (2.27) | 4.31 (2.27)
  Week 4: number analyzed (Participants) | 14 | 22 | 16 | 18 | 18
  Week 4 | 3.29 (2.46) | 3.45 (2.42) | 3.06 (2.35) | 3.67 (2.40) | 3.89 (2.63)
  Week 5: number analyzed (Participants) | 14 | 16 | 15 | 16 | 18
  Week 5 | 3.64 (2.37) | 4.56 (2.19) | 3.93 (2.66) | 3.25 (2.57) | 4.22 (2.53)
  Week 6: number analyzed (Participants) | 15 | 20 | 14 | 17 | 13
  Week 6 | 3.67 (2.32) | 3.25 (2.20) | 3.79 (2.22) | 3.06 (2.33) | 4.54 (2.60)
  Week 7: number analyzed (Participants) | 16 | 11 | 14 | 14 | 15
  Week 7 | 3.69 (2.30) | 5.00 (2.00) | 3.93 (2.37) | 3.50 (2.38) | 4.47 (2.36)
  Week 8: number analyzed (Participants) | 15 | 14 | 13 | 12 | 14
  Week 8 | 4.00 (2.07) | 4.57 (1.91) | 3.85 (2.58) | 3.58 (2.61) | 4.29 (2.05)
  Week 9: number analyzed (Participants) | 13 | 13 | 14 | 12 | 12
  Week 9 | 4.23 (1.74) | 4.62 (1.76) | 4.07 (2.37) | 4.08 (2.43) | 3.83 (2.37)
  Week 10: number analyzed (Participants) | 15 | 14 | 11 | 9 | 12
  Week 10 | 3.13 (1.92) | 3.71 (2.05) | 4.36 (2.46) | 4.22 (2.86) | 4.33 (2.46)
  Week 11: number analyzed (Participants) | 13 | 11 | 11 | 10 | 13
  Week 11 | 4.23 (2.24) | 4.00 (2.41) | 4.18 (2.32) | 3.90 (2.64) | 4.08 (2.60)
  Week 12: number analyzed (Participants) | 11 | 10 | 9 | 11 | 12
  Week 12 | 3.64 (2.01) | 4.60 (1.90) | 5.00 (2.50) | 4.09 (2.43) | 3.83 (2.41)
  Week 13: number analyzed (Participants) | 13 | 10 | 9 | 9 | 11
  Week 13 | 3.15 (2.08) | 4.30 (1.64) | 4.67 (2.83) | 4.78 (2.28) | 4.45 (2.21)
  Week 14: number analyzed (Participants) | 13 | 10 | 8 | 10 | 13
  Week 14 | 3.69 (2.46) | 3.80 (2.25) | 4.63 (2.07) | 4.30 (2.58) | 4.08 (2.36)
  Week 15: number analyzed (Participants) | 12 | 7 | 10 | 9 | 8
  Week 15 | 3.17 (2.17) | 4.00 (2.58) | 3.60 (2.59) | 3.33 (2.40) | 5.00 (2.00)
  Week 16: number analyzed (Participants) | 8 | 6 | 7 | 10 | 7
  Week 16 | 3.50 (1.93) | 4.67 (2.16) | 4.14 (1.95) | 3.90 (2.81) | 4.57 (1.27)
  Week 17: number analyzed (Participants) | 9 | 7 | 7 | 9 | 9
  Week 17 | 3.67 (2.45) | 3.29 (2.29) | 4.43 (2.15) | 3.44 (2.46) | 3.67 (2.18)
  Week 18: number analyzed (Participants) | 8 | 7 | 6 | 7 | 6
  Week 18 | 3.63 (2.00) | 3.29 (1.60) | 4.50 (1.64) | 3.14 (2.67) | 4.67 (2.42)
  Week 19: number analyzed (Participants) | 9 | 8 | 5 | 7 | 7
  Week 19 | 3.89 (2.37) | 2.50 (1.41) | 4.60 (2.51) | 3.71 (2.43) | 3.57 (2.57)
  Week 20: number analyzed (Participants) | 6 | 5 | 8 | 7 | 6
  Week 20 | 4.83 (1.72) | 3.20 (2.59) | 4.00 (2.39) | 3.29 (1.98) | 4.00 (2.37)
  Week 21: number analyzed (Participants) | 6 | 5 | 7 | 8 | 3
  Week 21 | 3.83 (2.40) | 3.40 (2.51) | 2.29 (1.38) | 2.38 (2.13) | 5.67 (1.53)
  Week 22: number analyzed (Participants) | 8 | 6 | 4 | 6 | 3
  Week 22 | 3.38 (1.69) | 3.17 (2.14) | 4.25 (2.75) | 3.17 (2.14) | 4.67 (3.21)
  Week 23: number analyzed (Participants) | 8 | 5 | 4 | 4 | 3
  Week 23 | 4.50 (2.07) | 3.60 (2.30) | 4.25 (2.06) | 2.75 (2.22) | 4.67 (3.21)
  Week 24: number analyzed (Participants) | 6 | 3 | 2 | 4 | 3
  Week 24 | 4.50 (2.51) | 4.00 (2.00) | 7.00 (0.00) | 3.25 (2.87) | 5.67 (2.31)

22. Secondary Outcome: Amount of Rescue Medication Taken Per Week
Description: In case of inadequate pain relief or worsening symptoms of IC/PBS, acetaminophen up to 3000 mg per day (1500 mg/day for Japanese population) could be taken as rescue medication.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 22 | 27 | 21 | 20 | 23
mg/week
  Baseline | 5827.3 (4485.87) | 4781.5 (4596.49) | 5428.6 (4688.51) | 5875.0 (4795.49) | 5695.7 (4255.32)
  Week 1: number analyzed (Participants) | 18 | 22 | 18 | 20 | 17
  Week 1 | 5527.8 (3908.78) | 5090.9 (4055.09) | 5444.4 (6125.86) | 6375.0 (4737.52) | 6058.8 (3273.39)
  Week 2: number analyzed (Participants) | 21 | 22 | 20 | 20 | 17
  Week 2 | 4333.3 (4749.56) | 4590.9 (4052.15) | 5300.0 (5795.64) | 5369.6 (5341.13) | 5647.1 (4018.57)
  Week 3: number analyzed (Participants) | 15 | 21 | 18 | 19 | 16
  Week 3 | 4573.3 (4831.66) | 4190.5 (3838.87) | 5861.1 (5232.27) | 5368.4 (4669.17) | 6218.8 (4837.25)
  Week 4: number analyzed (Participants) | 14 | 22 | 16 | 18 | 18
  Week 4 | 4371.4 (4431.60) | 4013.6 (4024.84) | 4312.5 (4003.64) | 5500.0 (5787.92) | 5194.4 (4765.50)
  Week 5: number analyzed (Participants) | 14 | 16 | 15 | 16 | 18
  Week 5 | 4342.9 (4300.22) | 5625.0 (4368.45) | 5866.7 (5569.26) | 4843.8 (5545.93) | 5694.4 (4902.40)
  Week 6: number analyzed (Participants) | 15 | 20 | 14 | 17 | 13
  Week 6 | 4873.3 (4005.08) | 3320.0 (2758.83) | 5178.6 (4846.12) | 4735.3 (6200.09) | 6500.0 (4267.12)
  Week 7: number analyzed (Participants) | 16 | 11 | 14 | 14 | 15
  Week 7 | 5181.3 (4803.36) | 6181.8 (3363.57) | 5392.9 (4637.55) | 4928.6 (5473.21) | 6500.0 (4263.63)
  Week 8: number analyzed (Participants) | 15 | 14 | 13 | 12 | 14
  Week 8 | 4740.0 (2844.74) | 6071.4 (4367.08) | 6307.7 (6223.40) | 5875.0 (6045.75) | 6428.6 (4807.27)
  Week 9: number analyzed (Participants) | 13 | 13 | 14 | 12 | 12
  Week 9 | 5238.5 (2722.91) | 6884.6 (5838.64) | 6464.3 (6203.18) | 6166.7 (6087.74) | 5958.3 (5565.55)
  Week 10: number analyzed (Participants) | 15 | 14 | 11 | 9 | 12
  Week 10 | 4266.7 (3272.54) | 4785.7 (4259.44) | 7181.8 (5934.11) | 6333.3 (6359.05) | 6916.7 (5418.12)
  Week 11: number analyzed (Participants) | 13 | 11 | 11 | 10 | 13
  Week 11 | 5538.5 (3078.57) | 5681.8 (5316.36) | 5500.0 (4398.86) | 5750.0 (5422.43) | 6807.7 (7084.43)
  Week 12: number analyzed (Participants) | 11 | 10 | 9 | 11 | 12
  Week 12 | 4954.5 (3791.14) | 6250.0 (5731.25) | 6333.3 (3848.70) | 7500.0 (7861.30) | 5583.3 (5142.66)
  Week 13: number analyzed (Participants) | 13 | 10 | 9 | 9 | 11
  Week 13 | 6500.0 (8638.58) | 5800.0 (4211.10) | 6777.8 (5810.07) | 6888.9 (6406.92) | 6772.7 (4808.14)
  Week 14: number analyzed (Participants) | 13 | 10 | 8 | 10 | 13
  Week 14 | 6269.2 (5666.48) | 5250.0 (4184.96) | 5562.5 (3310.56) | 6250.0 (6161.03) | 6807.7 (5717.44)
  Week 15: number analyzed (Participants) | 12 | 7 | 10 | 9 | 8
  Week 15 | 5083.3 (4655.56) | 8214.3 (8489.49) | 4700.0 (4601.93) | 7333.3 (8437.27) | 6500.0 (3909.69)
  Week 16: number analyzed (Participants) | 8 | 6 | 7 | 10 | 7
  Week 16 | 5375.0 (4332.19) | 6083.3 (3292.67) | 5500.0 (3807.89) | 6900.0 (6814.20) | 6142.9 (2925.67)
  Week 17: number analyzed (Participants) | 9 | 7 | 7 | 9 | 9
  Week 17 | 6000.0 (5454.36) | 3571.4 (3207.13) | 6000.0 (4133.20) | 4722.2 (3392.19) | 6111.1 (6303.66)
  Week 18: number analyzed (Participants) | 8 | 7 | 6 | 7 | 6
  Week 18 | 6437.5 (6038.20) | 3285.7 (2766.72) | 6583.3 (4128.16) | 3714.3 (3672.61) | 5583.3 (4079.42)
  Week 19: number analyzed (Participants) | 9 | 8 | 5 | 7 | 7
  Week 19 | 6500.0 (4242.64) | 4250.0 (4157.61) | 6400.0 (5042.32) | 4214.3 (3717.72) | 4214.3 (4270.61)
  Week 20: number analyzed (Participants) | 6 | 5 | 8 | 7 | 6
  Week 20 | 7333.3 (4191.26) | 3300.0 (3290.14) | 5375.0 (4413.86) | 3714.3 (3186.65) | 5000.0 (5167.20)
  Week 21: number analyzed (Participants) | 6 | 5 | 7 | 8 | 3
  Week 21 | 6333.3 (4792.36) | 3600.0 (3595.14) | 2428.6 (1592.39) | 2750.0 (2563.48) | 7333.3 (7333.3)
  Week 22: number analyzed (Participants) | 8 | 6 | 4 | 6 | 3
  Week 22 | 5625.0 (3482.10) | 2750.0 (2715.70) | 5375.0 (4534.59) | 5250.0 (3489.27) | 6000.0 (4582.58)
  Week 23: number analyzed (Participants) | 8 | 5 | 4 | 4 | 3
  Week 23 | 8375.0 (5566.16) | 3300.0 (2841.65) | 4500.0 (2886.75) | 3125.0 (1931.11) | 6666.7 (5507.57)
  Week 24: number analyzed (Participants) | 6 | 3 | 2 | 4 | 3
  Week 24 | 7500.0 (4560.70) | 3166.7 (2020.73) | 6000.0 (2121.32) | 3625.0 (2780.14) | 8500.0 (5766.28)

23. Secondary Outcome: Serum Total Nerve Growth Factor (NGF) Levels
Description: Serum samples were analyzed for total NGF using a validated, sensitive and specific immunoaffinity enrichment liquid chromatography tandem mass spectrometric method (IA/LC/MS/MS) method.
Time Frame: Baseline, Week 1, 2, 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 40 | 39 | 36 | 40 | 40
picogram per milliliter (pg/mL)
  Baseline: number analyzed (Participants) | 35 | 36 | 34 | 34 | 33
  Baseline | 41.756 (11.5576) | 39.929 (10.7855) | 37.209 (8.4699) | 38.381 (11.0441) | 38.150 (7.6355)
  Week 1 | 39.260 (13.2510) | 552.485 (221.4202) | 730.917 (253.8217) | 1034.317 (221.8687) | 1113.780 (307.0217)
  Week 2: number analyzed (Participants) | 37 | 37 | 34 | 36 | 34
  Week 2 | 40.162 (10.1141) | 901.633 (335.4488) | 1242.388 (425.2031) | 1644.283 (396.6413) | 1812.559 (530.0335)
  Week 8: number analyzed (Participants) | 35 | 34 | 27 | 30 | 31
  Week 8 | 58.075 (103.6542) | 841.984 (446.1437) | 1545.148 (770.2641) | 2502.127 (833.8403) | 3369.039 (1795.1505)
  Week 16: number analyzed (Participants) | 29 | 30 | 24 | 25 | 26
  Week 16 | 48.207 (28.6793) | 590.896 (638.2373) | 1079.050 (803.0958) | 3171.980 (1205.2251) | 3497.462 (2837.0678)
  Week 24: number analyzed (Participants) | 19 | 18 | 18 | 18 | 17
  Week 24 | 40.626 (8.9706) | 131.474 (123.8849) | 321.928 (331.1179) | 2153.000 (929.5347) | 3137.829 (3612.2725)

24. Other Pre Specified Outcome: Number of Participants With Neurological Examination Findings
Description: A neurological examination assessed the strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index fingers and great toes.
Time Frame: Week 2, 8, 16, Week 24 or early termination
Population: ITT analysis set. Here 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'number analyzed' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 39 | 39
Participants
  Week 2 | 1 | 4 | 1 | 5 | 0
  Week 8: number analyzed (Participants) | 34 | 35 | 28 | 29 | 31
  Week 8 | 2 | 2 | 0 | 3 | 1
  Week 16: number analyzed (Participants) | 22 | 10 | 19 | 20 | 19
  Week 16 | 0 | 1 | 2 | 4 | 1
  Week 24 or early termination: number analyzed (Participants) | 38 | 26 | 29 | 32 | 35
  Week 24 or early termination | 1 | 2 | 1 | 5 | 2

25. Other Pre Specified Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 2, 8, 16 and 24
Description: The NIS constituted the sum of 37 standard items of neuromuscular examination used to assess the muscle strength, reflexes and sensation. Each item was scored separately for left and right sides. Components of muscle weakness (24 items) were scored on a scale from 0 (normal) to 4 (paralysis), with higher score = more weakness; components of reflexes and sensation (13 items) scored on a scale with 0 = normal, 1 = decreased or 2 = absent. Total NIS score ranged from 0 to 244, a higher score indicate more impairment.
Time Frame: Baseline, Week 2, 8, 16, 24
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study medication. Here 'number analyzed' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
units on a scale
  Baseline | 1.0 (3.46) | 0.4 (0.92) | 0.9 (3.10) | 0.9 (2.87) | 0.3 (0.84)
  Change at Week 2: number analyzed (Participants) | 42 | 41 | 37 | 39 | 39
  Change at Week 2 | -0.7 (3.45) | 0.2 (0.86) | 0.2 (1.32) | 0.9 (2.88) | -0.0 (0.16)
  Change at Week 8: number analyzed (Participants) | 34 | 35 | 28 | 29 | 31
  Change at Week 8 | -0.5 (3.53) | 0.3 (1.38) | -0.1 (0.47) | 1.1 (5.28) | 0.0 (0.41)
  Change at Week 16: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Change at Week 16 | -0.1 (0.43) | -0.3 (0.66) | 0.3 (1.16) | 1.4 (6.33) | 0.1 (0.23)
  Change at Week 24: number analyzed (Participants) | 38 | 36 | 29 | 32 | 35
  Change at Week 24 | -0.4 (1.75) | -0.1 (0.63) | -0.6 (1.74) | 0.7 (5.15) | 0.1 (0.37)

26. Other Pre Specified Outcome: Body Temperature
Time Frame: Screening, Day 1 (1 hour pre-dose and post-dose), Week 1, 2, Week 8 (1 hour pre-dose and post-dose), Week 16, 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
degree Celsius
  Screening: number analyzed (Participants) | 42 | 39 | 37 | 40 | 39
  Screening | 36.56 (0.323) | 36.71 (0.304) | 36.56 (0.363) | 36.58 (0.341) | 36.67 (0.328)
  Day 1 (1 hour pre-dose): number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
  Day 1 (1 hour pre-dose) | 36.56 (0.359) | 36.62 (0.327) | 36.64 (0.321) | 36.55 (0.362) | 36.57 (0.246)
  Day 1 (1 hour post-dose): number analyzed (Participants) | 41 | 41 | 36 | 39 | 39
  Day 1 (1 hour post-dose) | 36.46 (0.306) | 36.55 (0.372) | 36.65 (0.304) | 36.50 (0.364) | 36.58 (0.322)
  Week 1 | 36.57 (0.338) | 36.67 (0.351) | 36.52 (0.349) | 36.58 (0.317) | 36.48 (0.351)
  Week 2: number analyzed (Participants) | 41 | 41 | 37 | 39 | 40
  Week 2 | 36.56 (0.397) | 36.57 (0.401) | 36.55 (0.376) | 36.63 (0.360) | 36.54 (0.294)
  Week 8 (1 hour pre-dose): number analyzed (Participants) | 34 | 35 | 27 | 29 | 31
  Week 8 (1 hour pre-dose) | 36.56 (0.321) | 36.59 (0.285) | 36.66 (0.342) | 36.58 (0.339) | 36.60 (0.350)
  Week 8 (1 hour post-dose): number analyzed (Participants) | 19 | 19 | 18 | 19 | 16
  Week 8 (1 hour post-dose) | 36.57 (0.307) | 36.63 (0.301) | 36.60 (0.350) | 36.45 (0.244) | 36.66 (0.305)
  Week 16: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Week 16 | 36.53 (0.353) | 36.66 (0.398) | 36.64 (0.341) | 36.37 (0.299) | 36.71 (0.251)
  Week 24: number analyzed (Participants) | 38 | 35 | 30 | 33 | 35
  Week 24 | 36.60 (0.387) | 36.63 (0.411) | 36.53 (0.368) | 36.53 (0.325) | 36.60 (0.300)

27. Other Pre Specified Outcome: Systolic and Diastolic Blood Pressure
Description: Systolic Blood Pressure (SBP) is the blood pressure (pressure exerted by circulating blood on the walls of blood vessels) when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle of heart. Diastolic Blood Pressure (DBP) is the blood pressure (pressure exerted by circulating blood on the walls of blood vessels) when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles of heart.
Time Frame: Screening, Day 1 (1 hour pre-dose and post-dose), Week 1, 2, Week 8 (1 hour pre-dose and post-dose), Week 16, 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
millimeter of mercury (mmHg)
  Screening: SBP | 126.3 (15.95) | 118.5 (14.15) | 121.3 (12.25) | 123.5 (12.40) | 123.2 (13.39)
  Screening: DBP | 75.4 (11.46) | 73.4 (9.05) | 76.4 (9.46) | 76.8 (10.35) | 75.0 (9.34)
  Day 1 (1 hour pre-dose): SBP | 125.8 (16.81) | 118.0 (13.88) | 119.4 (12.02) | 121.1 (14.86) | 121.3 (12.75)
  Day 1 (1 hour pre-dose): DBP | 75.9 (10.13) | 73.1 (8.60) | 75.9 (10.61) | 74.5 (10.02) | 75.5 (9.47)
  Day 1(1 hour post-dose): SBP | 125.0 (13.06) | 118.5 (12.41) | 121.5 (12.78) | 123.4 (15.02) | 122.7 (14.17)
  Day 1(1 hour post-dose): DBP | 74.2 (9.41) | 74.5 (8.77) | 73.8 (11.72) | 74.8 (9.05) | 76.8 (8.65)
  Week 1: SBP | 124.6 (17.29) | 117.4 (14.44) | 116.8 (12.07) | 117.9 (13.35) | 119.4 (12.44)
  Week 1: DBP | 74.9 (11.27) | 72.6 (9.42) | 74.7 (9.69) | 71.6 (9.88) | 73.9 (10.32)
  Week 2: SBP: number analyzed (Participants) | 42 | 41 | 37 | 39 | 40
  Week 2: SBP | 124.4 (14.26) | 113.3 (11.82) | 118.8 (13.47) | 122.0 (16.45) | 118.2 (12.53)
  Week 2: DBP: number analyzed (Participants) | 42 | 41 | 37 | 39 | 40
  Week 2: DBP | 74.8 (8.85) | 71.3 (8.46) | 76.8 (8.99) | 74.5 (9.44) | 72.4 (9.15)
  Week 8(1 hour pre-dose): SBP: number analyzed (Participants) | 34 | 35 | 28 | 29 | 31
  Week 8(1 hour pre-dose): SBP | 120.1 (12.64) | 115.1 (13.42) | 117.0 (14.06) | 122.4 (17.13) | 113.4 (11.83)
  Week 8(1 hour pre-dose): DBP: number analyzed (Participants) | 34 | 35 | 28 | 29 | 31
  Week 8(1 hour pre-dose): DBP | 73.8 (9.07) | 73.5 (9.93) | 72.0 (7.08) | 73.4 (9.73) | 71.5 (7.98)
  Week 8(1 hour post-dose): SBP: number analyzed (Participants) | 20 | 19 | 19 | 20 | 17
  Week 8(1 hour post-dose): SBP | 123.0 (12.39) | 111.8 (11.12) | 119.1 (9.18) | 120.7 (17.35) | 118.8 (9.98)
  Week 8(1 hour post-dose): DBP: number analyzed (Participants) | 20 | 19 | 19 | 20 | 17
  Week 8(1 hour post-dose): DBP | 73.9 (7.71) | 69.9 (8.63) | 75.2 (6.07) | 74.8 (9.34) | 73.8 (6.15)
  Week 16: SBP: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Week 16: SBP | 125.4 (17.72) | 117.4 (13.72) | 119.7 (13.63) | 121.8 (14.89) | 115.8 (10.33)
  Week 16: DBP: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Week 16: DBP | 75.3 (10.51) | 71.2 (8.24) | 72.8 (12.69) | 75.7 (12.15) | 71.2 (9.94)
  Week 24: SBP: number analyzed (Participants) | 37 | 35 | 29 | 33 | 35
  Week 24: SBP | 124.3 (16.37) | 118.3 (12.06) | 122.1 (12.78) | 122.4 (17.38) | 120.0 (12.43)
  Week 24: DBP: number analyzed (Participants) | 37 | 35 | 29 | 33 | 35
  Week 24: DBP | 77.6 (9.66) | 71.9 (10.13) | 78.1 (8.58) | 73.8 (10.05) | 74.1 (7.70)

28. Other Pre Specified Outcome: Heart Rate
Time Frame: Screening, Day 1 (1 hour pre-dose and post-dose), Week 1, 2, Week 8 (1 hour pre-dose and post-dose), Week 16, 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
beats per minute
  Screening | 74.7 (10.37) | 76.4 (10.40) | 75.0 (12.72) | 74.2 (15.22) | 75.5 (11.81)
  Day 1 (1 hour pre-dose): number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
  Day 1 (1 hour pre-dose) | 75.4 (10.45) | 77.5 (10.86) | 75.5 (12.06) | 73.6 (14.03) | 76.5 (11.17)
  Day 1 (1 hour post-dose): number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
  Day 1 (1 hour post-dose) | 75.1 (10.22) | 75.3 (9.18) | 74.8 (12.30) | 71.9 (12.76) | 75.3 (10.60)
  Week 1 | 77.2 (10.66) | 79.4 (11.07) | 76.4 (12.06) | 72.4 (14.00) | 80.1 (12.74)
  Week 2: number analyzed (Participants) | 42 | 41 | 37 | 39 | 40
  Week 2 | 76.1 (11.24) | 77.1 (10.36) | 75.8 (10.92) | 74.0 (14.22) | 77.8 (11.37)
  Week 8 (1 hour pre-dose): number analyzed (Participants) | 34 | 35 | 28 | 29 | 31
  Week 8 (1 hour pre-dose) | 74.7 (10.91) | 77.4 (14.51) | 71.1 (10.43) | 71.4 (15.02) | 75.1 (11.34)
  Week 8 (1 hour post-dose): number analyzed (Participants) | 20 | 19 | 19 | 20 | 17
  Week 8 (1 hour post-dose) | 73.9 (9.59) | 77.3 (12.66) | 72.3 (10.92) | 69.2 (15.58) | 71.3 (11.29)
  Week 16: number analyzed (Participants) | 22 | 20 | 18 | 20 | 19
  Week 16 | 75.6 (9.84) | 75.0 (11.54) | 75.9 (11.95) | 70.9 (15.77) | 75.6 (13.60)
  Week 24: number analyzed (Participants) | 38 | 35 | 30 | 33 | 35
  Week 24 | 77.5 (10.44) | 79.9 (11.68) | 75.3 (11.22) | 72.7 (13.81) | 77.3 (9.65)

29. Other Pre Specified Outcome: Respiratory Rate
Time Frame: Screening, Day 1 (1 hour pre-dose and post-dose), Week 1, 2, Week 8 (1 hour pre-dose and post-dose), Week 16, 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
respirations per minute
  Screening: number analyzed (Participants) | 42 | 41 | 37 | 40 | 39
  Screening | 16.2 (2.46) | 15.8 (2.89) | 16.3 (1.74) | 16.5 (2.83) | 16.1 (1.75)
  Day 1 (1 hour pre-dose) | 16.3 (2.62) | 16.2 (2.35) | 15.9 (2.14) | 16.2 (2.97) | 15.9 (1.83)
  Day 1 (1 hour post-dose) | 16.2 (2.64) | 16.3 (2.46) | 15.8 (2.42) | 16.2 (3.04) | 15.8 (1.98)
  Week 1 | 16.3 (2.64) | 16.3 (2.33) | 16.1 (2.08) | 16.2 (2.99) | 15.7 (2.09)
  Week 2: number analyzed (Participants) | 41 | 41 | 37 | 39 | 40
  Week 2 | 16.0 (2.49) | 16.4 (2.31) | 16.2 (2.29) | 16.8 (2.77) | 16.2 (1.94)
  Week 8 (1 hour pre-dose): number analyzed (Participants) | 34 | 35 | 27 | 29 | 31
  Week 8 (1 hour pre-dose) | 15.8 (2.75) | 15.8 (2.19) | 16.3 (2.25) | 15.9 (3.02) | 16.1 (1.88)
  Week 8 (1 hour post-dose): number analyzed (Participants) | 20 | 19 | 19 | 20 | 17
  Week 8 (1 hour post-dose) | 16.2 (2.89) | 16.3 (2.18) | 16.6 (1.87) | 16.4 (3.00) | 16.0 (1.54)
  Week 16: number analyzed (Participants) | 21 | 20 | 19 | 20 | 19
  Week 16 | 16.0 (2.00) | 16.9 (2.38) | 17.0 (2.24) | 16.2 (2.56) | 16.0 (1.67)
  Week 24: number analyzed (Participants) | 35 | 35 | 28 | 33 | 35
  Week 24 | 16.1 (2.67) | 15.6 (2.38) | 15.1 (2.40) | 16.0 (2.64) | 15.8 (2.08)

30. Other Pre Specified Outcome: Electrocardiogram Parameters: RR, PR, QRS, QT and Corrected QT (QTcB and QTcF) Intervals
Description: Following parameters were analyzed for ECG: RR interval, PR interval, QRS complex, QT interval, QT interval corrected using the Fridericia formula (QTcF), and QT interval corrected using the Bazett's formula (QTcB).
Time Frame: Screening, Day 1, Week 2, 8, 16, 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
millisecond (msec)
  Screening: RR Interval | 868.9 (152.10) | 863.3 (138.89) | 849.6 (136.23) | 878.5 (189.33) | 863.2 (143.31)
  Screening: PR Interval: number analyzed (Participants) | 42 | 41 | 37 | 38 | 40
  Screening: PR Interval | 155.1 (22.47) | 154.3 (19.60) | 156.4 (20.83) | 154.8 (24.53) | 158.6 (28.85)
  Screening: QRS Complex: number analyzed (Participants) | 42 | 41 | 37 | 39 | 40
  Screening: QRS Complex | 90.2 (7.23) | 89.0 (11.62) | 88.6 (8.33) | 87.5 (9.17) | 90.6 (6.82)
  Screening: QT Interval: number analyzed (Participants) | 42 | 40 | 37 | 38 | 40
  Screening: QT Interval | 389.1 (26.58) | 386.0 (28.24) | 389.1 (27.69) | 390.5 (37.31) | 384.0 (29.36)
  Screening: QTcB Interval: number analyzed (Participants) | 42 | 40 | 37 | 38 | 40
  Screening: QTcB Interval | 420.2 (24.73) | 418.0 (20.17) | 424.2 (22.27) | 416.8 (22.81) | 415.3 (19.71)
  Screening: QTcF Interval: number analyzed (Participants) | 42 | 40 | 37 | 38 | 40
  Screening: QTcF Interval | 409.3 (19.44) | 406.8 (18.29) | 411.9 (19.10) | 407.3 (21.13) | 404.3 (17.83)
  Day 1: RR Interval: number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
  Day 1: RR Interval | 852.3 (149.92) | 848.7 (137.85) | 849.4 (126.73) | 883.4 (183.93) | 836.4 (117.33)
  Day 1: PR Interval: number analyzed (Participants) | 40 | 41 | 37 | 37 | 39
  Day 1: PR Interval | 153.9 (20.71) | 156.1 (17.76) | 153.6 (22.14) | 153.2 (23.98) | 158.2 (34.39)
  Day 1: QRS Complex: number analyzed (Participants) | 41 | 41 | 37 | 39 | 40
  Day 1: QRS Complex | 87.6 (8.43) | 90.2 (9.91) | 87.3 (8.34) | 87.4 (10.46) | 89.1 (8.13)
  Day 1: QT Interval: number analyzed (Participants) | 40 | 38 | 37 | 39 | 39
  Day 1: QT Interval | 391.4 (31.92) | 382.1 (33.15) | 386.2 (27.28) | 392.5 (33.74) | 382.8 (23.82)
  Day 1: QTcB Interval: number analyzed (Participants) | 40 | 38 | 37 | 39 | 39
  Day 1: QTcB Interval | 425.6 (21.20) | 416.9 (18.02) | 420.8 (20.52) | 418.9 (18.21) | 418.4 (17.21)
  Day 1: QTcF Interval: number analyzed (Participants) | 40 | 38 | 37 | 39 | 39
  Day 1: QTcF Interval | 413.6 (19.16) | 404.8 (19.19) | 408.7 (18.27) | 409.5 (15.95) | 406.0 (15.28)
  Week 2: RR Interval: number analyzed (Participants) | 42 | 41 | 36 | 39 | 40
  Week 2: RR Interval | 835.3 (140.48) | 825.1 (117.52) | 857.5 (123.18) | 867.4 (191.34) | 833.4 (134.21)
  Week 2: PR Interval: number analyzed (Participants) | 42 | 41 | 36 | 38 | 40
  Week 2: PR Interval | 151.1 (21.46) | 158.4 (20.83) | 158.9 (21.31) | 152.7 (24.00) | 160.8 (28.15)
  Week 2: QRS Complex: number analyzed (Participants) | 42 | 41 | 36 | 39 | 40
  Week 2: QRS Complex | 88.5 (8.81) | 89.6 (12.50) | 89.6 (9.51) | 88.5 (8.50) | 90.0 (7.07)
  Week 2: QT Interval: number analyzed (Participants) | 41 | 40 | 36 | 39 | 40
  Week 2: QT Interval | 382.6 (27.92) | 382.6 (30.00) | 389.5 (29.46) | 386.4 (36.77) | 382.0 (23.45)
  Week 2: QTcB Interval: number analyzed (Participants) | 41 | 40 | 36 | 39 | 40
  Week 2: QTcB Interval | 422.6 (23.99) | 423.1 (21.21) | 422.1 (17.73) | 418.1 (20.29) | 420.9 (20.48)
  Week 2: QTcF Interval: number analyzed (Participants) | 41 | 40 | 36 | 39 | 40
  Week 2: QTcF Interval | 408.6 (19.88) | 408.9 (20.89) | 410.6 (17.61) | 406.7 (18.85) | 407.3 (15.44)
  Week 8: RR Interval: number analyzed (Participants) | 34 | 34 | 28 | 29 | 31
  Week 8: RR Interval | 849.6 (134.00) | 842.7 (121.90) | 855.0 (126.13) | 919.6 (199.85) | 882.8 (152.53)
  Week 8: PR Interval: number analyzed (Participants) | 33 | 32 | 28 | 27 | 30
  Week 8: PR Interval | 153.4 (20.12) | 158.6 (19.44) | 157.0 (22.20) | 154.3 (25.04) | 156.8 (29.74)
  Week 8: QRS Complex: number analyzed (Participants) | 34 | 34 | 28 | 29 | 31
  Week 8: QRS Complex | 87.4 (9.88) | 88.1 (11.59) | 89.4 (9.69) | 88.7 (10.52) | 90.5 (7.80)
  Week 8: QT Interval: number analyzed (Participants) | 33 | 32 | 28 | 28 | 31
  Week 8: QT Interval | 385.8 (29.34) | 379.8 (30.21) | 387.3 (21.80) | 401.5 (40.44) | 392.0 (28.49)
  Week 8: QTcB Interval: number analyzed (Participants) | 33 | 32 | 28 | 28 | 31
  Week 8: QTcB Interval | 419.8 (21.38) | 414.7 (16.98) | 421.1 (24.04) | 419.3 (16.86) | 419.8 (20.18)
  Week 8: QTcF Interval: number analyzed (Participants) | 33 | 32 | 28 | 28 | 31
  Week 8: QTcF Interval | 407.8 (19.36) | 402.5 (18.11) | 409.2 (18.95) | 412.8 (18.30) | 410.0 (16.65)
  Week 16: RR Interval: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Week 16: RR Interval | 825.7 (109.43) | 847.5 (138.15) | 799.6 (87.02) | 925.9 (224.34) | 865.4 (188.59)
  Week 16: PR Interval: number analyzed (Participants) | 22 | 18 | 19 | 17 | 19
  Week 16: PR Interval | 152.1 (24.39) | 157.1 (17.66) | 155.2 (18.75) | 156.6 (26.49) | 150.5 (21.33)
  Week 16: QRS Complex: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Week 16: QRS Complex | 90.1 (7.69) | 89.3 (8.68) | 90.8 (8.85) | 89.2 (8.79) | 90.4 (6.33)
  Week 16: QT Interval: number analyzed (Participants) | 22 | 16 | 19 | 19 | 19
  Week 16: QT Interval | 386.6 (25.90) | 380.7 (35.74) | 381.3 (23.89) | 403.9 (37.73) | 385.8 (30.81)
  Week 16: QTcB Interval: number analyzed (Participants) | 22 | 16 | 19 | 19 | 19
  Week 16: QTcB Interval | 426.8 (20.63) | 418.0 (14.16) | 427.6 (25.18) | 421.6 (21.94) | 418.7 (24.51)
  Week 16: QTcF Interval: number analyzed (Participants) | 22 | 16 | 19 | 19 | 19
  Week 16: QTcF Interval | 412.8 (18.96) | 404.8 (17.65) | 411.4 (22.01) | 414.9 (17.40) | 406.9 (17.80)
  Week 24: RR Interval: number analyzed (Participants) | 38 | 36 | 30 | 33 | 35
  Week 24: RR Interval | 849.1 (116.70) | 850.6 (136.92) | 821.8 (122.24) | 894.9 (164.80) | 851.2 (106.90)
  Week 24: PR Interval: number analyzed (Participants) | 37 | 35 | 30 | 30 | 33
  Week 24: PR Interval | 155.4 (20.29) | 157.0 (17.56) | 157.7 (21.18) | 158.9 (23.25) | 159.1 (27.92)
  Week 24: QRS Complex: number analyzed (Participants) | 38 | 36 | 30 | 33 | 33
  Week 24: QRS Complex | 89.2 (7.68) | 87.2 (11.48) | 89.4 (8.10) | 88.9 (8.56) | 89.4 (7.77)
  Week 24: QT Interval: number analyzed (Participants) | 38 | 34 | 29 | 32 | 33
  Week 24: QT Interval | 384.7 (28.57) | 386.4 (34.67) | 388.3 (27.18) | 395.0 (33.83) | 383.5 (24.31)
  Week 24: QTcB Interval: number analyzed (Participants) | 38 | 34 | 29 | 32 | 33
  Week 24: QTcB Interval | 418.7 (19.71) | 418.7 (19.47) | 427.7 (21.73) | 419.5 (23.12) | 418.4 (19.80)
  Week 24: QTcF Interval: number analyzed (Participants) | 38 | 34 | 29 | 32 | 33
  Week 24: QTcF Interval | 406.8 (19.45) | 407.3 (21.52) | 413.9 (20.07) | 410.8 (20.48) | 406.3 (18.21)

31. Other Pre Specified Outcome: Electrocardiogram Parameter: Heart Rate
Time Frame: Screening, Day 1, Week 2, 8, 16, 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
beats per minute
  Screening | 71.1 (12.18) | 71.2 (10.77) | 72.4 (11.49) | 71.3 (14.47) | 71.4 (12.42)
  Day 1: number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
  Day 1 | 72.4 (12.41) | 72.5 (11.34) | 72.3 (11.58) | 70.7 (14.36) | 73.2 (11.06)
  Week 2: number analyzed (Participants) | 42 | 41 | 36 | 39 | 40
  Week 2 | 73.9 (12.46) | 74.1 (10.38) | 71.5 (10.94) | 72.0 (13.98) | 73.8 (11.68)
  Week 8: number analyzed (Participants) | 34 | 34 | 28 | 29 | 31
  Week 8 | 72.3 (11.47) | 72.8 (11.66) | 71.7 (10.93) | 68.4 (15.47) | 69.9 (12.56)
  Week 16: number analyzed (Participants) | 22 | 20 | 19 | 20 | 19
  Week 16 | 73.8 (9.77) | 72.9 (12.76) | 75.9 (8.69) | 68.3 (15.39) | 72.2 (14.41)
  Week 24: number analyzed (Participants) | 38 | 36 | 30 | 33 | 35
  Week 24 | 71.9 (9.81) | 72.4 (11.98) | 74.7 (11.55) | 69.3 (13.12) | 71.5 (9.09)

32. Other Pre Specified Outcome: Post-void Residual (PVR) Volume
Description: PVR volume is an objective assessment of the amount of urine left in the bladder after normal urination and will monitor whether the active treatment is having an adverse effect on lower urinary tract voiding function. The PVR volume assessed using trans-abdominal ultrasound (e.g., bladder scanner) with the participant in a supine position immediately after voluntary urination.
Time Frame: Screening, Week 2, 8, 16, 24
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study medication. Here 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure. 'number analyzed' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 39 | 40
milliliter
  Screening: number analyzed (Participants) | 41 | 41 | 37 | 39 | 40
  Screening | 27.1 (31.44) | 22.3 (33.29) | 24.8 (36.99) | 25.2 (27.10) | 24.5 (35.56)
  Week 2 | 20.9 (30.43) | 11.6 (17.16) | 20.1 (34.58) | 20.7 (28.03) | 25.8 (39.61)
  Week 8: number analyzed (Participants) | 32 | 33 | 28 | 27 | 30
  Week 8 | 19.2 (24.37) | 11.9 (21.47) | 17.7 (21.36) | 21.4 (32.82) | 21.2 (29.39)
  Week 16: number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
  Week 16 | 20.5 (37.61) | 10.9 (15.33) | 27.3 (47.43) | 25.7 (26.40) | 23.9 (31.41)
  Week 24: number analyzed (Participants) | 38 | 34 | 30 | 31 | 35
  Week 24 | 17.2 (25.05) | 14.3 (24.27) | 18.6 (33.84) | 16.8 (25.50) | 17.6 (22.14)

33. Other Pre Specified Outcome: Number of Participants With Urinalysis Abnormalities
Description: Urine was tested for specific gravity, pH, protein, glucose, ketones, blood, bilirubin, nitrites, and leukocyte, esterase using a urine dipstick. Number of participants with a laboratory abnormality meeting specified criteria: specific gravity (<1.003 and >1.030), urine pH (<4.5 and >8), protein (>=1 value in qualitative test), glucose (>=1 value in qualitative test), ketones (>=1 value in qualitative test), blood (>=1 value in qualitative test), bilirubin (>=1 value in qualitative test), nitrites (>=1), and leukocyte esterase (>=1) are reported.
Time Frame: Screening up to Week 24
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 40 | 41 | 37 | 40 | 40
Participants
  Urine Specific Gravity: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Urine Specific Gravity |  |  |  |  | 0
  Urine pH | 1 | 0 | 0 | 1 | 0
  Urine Glucose | 0 | 1 | 0 | 0 | 1
  Urine Ketones | 1 | 3 | 2 | 0 | 4
  Urine Protein | 3 | 1 | 2 | 0 | 5
  Urine Blood | 10 | 11 | 8 | 11 | 10
  Urine Bilirubin | 1 | 3 | 7 | 5 | 4
  Urine Nitrite | 1 | 0 | 1 | 0 | 2
  Urine Leukocyte Esterase | 3 | 4 | 3 | 6 | 3

34. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory examination included hematology, liver function, renal function, lipids, electrolytes, clinical chemistry, and urinalysis. Reported results include abnormal laboratory findings without regard to baseline abnormality.
Time Frame: Screening up to Week 24
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 41 | 41 | 37 | 40 | 40
Participants | 28 | 21 | 24 | 24 | 25

35. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to 112 days after the last dose (up to Week 24)
Population: Safety analysis set included all randomized participants who had received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 42 | 41 | 37 | 40 | 40
Participants
  AEs | 24 | 30 | 24 | 29 | 23
  SAEs | 0 | 4 | 6 | 1 | 1

36. Other Pre Specified Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA). In this outcome measure number of participants with presence of anti-tanezumab antibodies are reported.
Time Frame: Baseline, Week 8, 16, 24
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Number analyzed (Participants) | 36 | 33 | 35 | 36
Participants
  Baseline | 0 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 34 | 27 | 30 | 30
  Week 8 | 0 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 30 | 24 | 25 | 26
  Week 16 | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 18 | 18 | 17 | 17
  Week 24 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Any clinical significant changes in physical examination and vital sign findings were reported as AEs.
Arm/Group | Placebo | Tanezumab 1 mg | Tanezumab 2.5 mg | Tanezumab 10 mg | Tanezumab 20 mg
Serious Adverse Events (participants affected / at risk) | 0/42 | 4/41 | 6/37 | 1/40 | 1/40
Other Adverse Events (participants affected / at risk) | 21/42 | 25/41 | 15/37 | 27/40 | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | Tanezumab 1 mg (N=41) | Tanezumab 2.5 mg (N=37) | Tanezumab 10 mg (N=40) | Tanezumab 20 mg (N=40)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | Tanezumab 1 mg (N=41) | Tanezumab 2.5 mg (N=37) | Tanezumab 10 mg (N=40) | Tanezumab 20 mg (N=40)
Eye swelling (Eye disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 1 | 2 | 1
Chest pain (General disorders) | 0 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 2 | 0 | 1
Injection site reaction (General disorders) | 4 | 4 | 0 | 2 | 2
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 6 | 1 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 3 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Decreased vibratory sense (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 3 | 0
Headache (Nervous system disorders) | 4 | 7 | 3 | 7 | 4
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 3 | 1
Paraesthesia (Nervous system disorders) | 3 | 3 | 0 | 9 | 2
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1 | 2 | 4 | 0
Cystitis interstitial (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of efficacy of all doses of tanezumab demonstrated during pre-planned interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.